# **Signature Page**

# Randomized Trial of Full-Time Occlusion Therapy for Intermittent Exotropia in Children

Funded by: The National Eye Institute of the National Institutes of Health

**Protocol Identifying Number: IXT7** 

Version Number: 1.0

19 April 2022

| Protocol Co-Chair | |
|---|---|
| Name, degree | Stephen P. Christiansen, MD |
| Title | Protocol Co-Chair |
| Institution Name | Department of Ophthalmology Boston Medical Center, Boston University School of Medicine 85 East Concord St, 8th Fl Boston, MA 02116 Phone: 617-638-4589 Cell: 617-735-5688 Email:Stephen.Christiansen@bmc.org |
| Signature/ Date | |
| Protocol Co-Chair | |
| Name, degree | Erin C Jenewein, OD, MS, FAAO |
| Title | Protocol Co-Chair |
| Institution Name | The Eye Institute 1200 West Godfrey Philadelphia, PA 19141 Cell: 920-456-9105 Email: ejenewein@salus.edu |
| Signature/ Date | |
| JCHR Lead Investigator | |
| Name, degree | Raymond T. Kraker, M.S.P.H. |
| Title | Principal Investigator, PEDIG Director |
| Institution Name | Jaeb Center for Health Research 15310 Amberly Drive, Suite 350 Tampa, FL 33647 Phone: 1-888-797-3344 Fax: 1-888-697-3344 Email: rkraker@jaeb.org |
| Signature/ Date | |

# Randomized Trial of Full-Time Occlusion Therapy for Intermittent Exotropia in Children

Funded by: The National Eye Institute of the National Institutes of Health

Protocol Identifying Number: IXT7 Version Number: 1.0

19 April 2022

IXT7ProtV1.0\_19Apr2022 

# **KEY ROLES**

| Protocol Co-Chair | |
|---|---|
| Name, degree | Stephen P. Christiansen, MD |
| Title | Protocol Co-Chair |
| Institution Name | Department of Ophthalmology Boston Medical Center, Boston University School of Medicine 85 East Concord St, 8th Fl Boston, MA 02116 Phone: 617-638-4589 Cell: 617-735-5688 Email:Stephen.Christiansen@bmc.org |
| Protocol Co-Chair | |
| Name, degree | Erin C Jenewein, OD, MS, FAAO |
| Title | Protocol Co-Chair |
| Institution Name | The Eye Institute 1200 West Godfrey Philadelphia, PA 19141 Cell: 920-456-9105 Email: ejenewein@salus.edu |
| JCHR Lead Investigator | |
| Name, degree | Raymond T. Kraker, M.S.P.H. |
| Title | Principal Investigator, PEDIG Director |
| Institution Name | Jaeb Center for Health Research 15310 Amberly Drive, Suite 350 Tampa, FL 33647 Phone: 1-888-797-3344 Fax: 1-888-697-3344 Email: rkraker@jaeb.org |

IXT7ProtV1.0\_19Apr2022 

# **TABLE OF CONTENTS**

| CHAPTER 1: BACKGROUND INFORMATION | 14 |
|---------------------------------------------------------------|----|
| 1.1 Epidemiology and Clinical Characteristics | 14 |
| 1.2 Current Management Strategies | 14 |
| 1.2.1 Observation | 14 |
| 1.2.2 Surgery | 15 |
| 1.2.3 Nonsurgical treatments | 15 |
| 1.3 Patching | 16 |
| 1.3.1 Current clinical practice | 16 |
| 1.3.2 Previous Randomized Trials of Patching Treatment | 16 |
| 1.3.3 Previous Non-randomized Studies of Patching Treatment | 17 |
| 1.4 Mechanism of Patching Treatment Effect | 18 |
| 1.4.1 Suppression | 18 |
| 1.4.2 Fusional Vergence Amplitudes | 18 |
| 1.4.3 Magnitude of Deviation | 18 |
| 1.5 Measuring Patch Wear Time | 18 |
| 1.6 Unanswered Questions Regarding Patching Treatment for IXT | 19 |
| 1.7 Rationale for Present Study | 19 |
| 1.8 Study Objectives | 19 |
| 1.9 Potential Risks and Benefits of Study Treatment | 20 |
| 1.9.1 Known Potential Risks | 20 |
| 1.9.2 Known Potential Benefits | 20 |
| 1.10 Risks of Examination or Testing Procedures | 20 |
| 1.11 Risk Assessment | 20 |
| 1.12 General Considerations | 20 |
| CHAPTER 2: STUDY ENROLLMENT AND RANDOMIZATION | |
| 2.1 Participant Recruitment and Enrollment | 21 |
| 2.1.1 Informed Consent | 21 |
| 2.2 Eligibility Criteria | 21 |
| 2.2.1 Inclusion Criteria | 21 |
| 2.2.2 Exclusion Criteria | |
| 2.3 Historical Information | 23 |
| 2.4 Screening and Baseline Procedures | 23 |
| 2.5 Randomization | 25 |
| 2.5.1 Observation Group | 25 |
| 2.5.2 Full-Time Patching Group | 25 |

| 2.6 Monitoring of Adherence | 25 |
|---------------------------------------------------------------|----|
| CHAPTER 3: STUDY FOLLOW-UP | 26 |
| 3.1 Study Visits | 26 |
| 3.2 Phone Call at 4-weeks | 26 |
| 3.3 Masking Procedures | 26 |
| 3.3.1 Masked Examiner | 26 |
| 3.4 Testing Procedures at 3-Month Outcome Visit | 26 |
| 3.5 IXT Treatment Changes During Follow-up | 27 |
| 3.6 Management of Refractive Error During Follow-up | 27 |
| CHAPTER 4: TESTING PROCEDURES AND QUESTIONNAIRES | 29 |
| 4.1 Clinical Assessments | 29 |
| CHAPTER 5: UNANTICIPATED PROBLEM AND ADVERSE EVENT REPORTING | 33 |
| 5.1 Unanticipated Problems. | 33 |
| 5.2 Adverse Events | 33 |
| 5.3 Safety Oversight | 33 |
| 5.4 Stopping Criteria | 34 |
| 5.5 Participant Discontinuation of Study Treatment | 34 |
| CHAPTER 6: MISCELLANEOUS CONSIDERATIONS | 35 |
| 6.1 Contacts by the Jaeb Center for Health Research and Sites | 35 |
| 6.2 Participant Compensation | 35 |
| 6.3 Participant Withdrawal | 35 |
| 6.4 Confidentiality | 35 |
| CHAPTER 7: STATISTICAL CONSIDERATIONS | 36 |
| 7.1 Statistical and Analytical Plans | 36 |
| 7.2 Primary Objective and Hypothesis | 36 |
| 7.3 Sample Size | 36 |
| 7.4 Interim Monitoring | 38 |
| 7.5 Analysis Datasets | 38 |
| 7.6 Analysis of the Primary Efficacy Endpoints | 38 |
| 7.6.1 Sensitivity Analyses | 39 |
| 7.7 Analysis of the Secondary Endpoints | 39 |
| 7.7.1 Near Control | 39 |
| 7.7.2 Angle of Deviation | 40 |
| 7.7.3 Level of Suppression | 40 |
| 7.7.4 Proportion with Anomalous Retinal Correspondence | 40 |

| 7.7.5 Convergence and Divergence Fusional Amplitudes | 40 |
|------------------------------------------------------|----|
| 7.7.6 IXT Symptom Survey Score | 40 |
| 7.7.7 PedEyeQ Score | 40 |
| 7.7.8 Binocular Diplopia by Parental Report | 40 |
| 7.8 Exploratory Analyses | 41 |
| 7.8.1 Actual Patch Wear Time | 41 |
| 7.8.2 Outcome of Retinal Correspondence Testing | 41 |
| 7.8.3 Subgroup Analysis of Distance Control | 42 |
| 7.9 Safety Analyses | 42 |
| 7.9.1 Deterioration | 42 |
| 7.9.2 Reduction of Distance Visual Acuity | 42 |
| 7.9.3 Diplopia | 42 |
| 7.10 Patching Adherence | 42 |
| 7.11 Additional Tabulations and Analyses | 42 |
| CHAPTER 8: DATA COLLECTION AND MONITORING | 43 |
| 8.1 Case Report Forms and Other Data Collection | |
| 8.2 Study Records Retention | 43 |
| 8.3 Quality Assurance and Monitoring | 43 |
| 8.4 Protocol Deviations | 44 |
| CHAPTER 9: ETHICS/PROTECTION OF HUMAN PARTICIPANTS | 45 |
| 9.1 Ethical Standard | 45 |
| 9.2 Institutional Review Boards | 45 |
| 9.3 Informed Consent Process | 45 |
| 9.3.1 Consent Procedures and Documentation | 45 |
| 9.3.2 Participant and Data Confidentiality | 45 |
| 9.3.3 Future Use of Data | 46 |
| Chapted 10. References | 47 |

# **LIST OF ABBREVIATIONS**

| ABBREVIATION | DEFINITION |
|---|---|
| Δ | Prism diopters |
| ANCOVA | Analysis of covariance |
| ATS | Amblyopia Treatment Study |
| ATS-HOTV | Amblyopia Treatment Study HOTV visual acuity testing protocol |
| CI | Confidence interval |
| CFR | Code of Federal Regulations |
| CR | Cycloplegic refraction |
| CRF | Case report form |
| D | Diopter |
| DHHS | Department of Health and Human Services |
| DSMC | Data safety and monitoring committee |
| eCRF | Electronic case report form |
| E-ETDRS | Electronic Early Treatment of Diabetic Retinopathy Study visual acuity protocol |
| EVA | Electronic visual acuity tester |
| FDA | Food and Drug Administration |
| FDR | False discovery rate |
| FT | Full-time patching |
| GCP | Good clinical practice |
| ICH | International Council for Harmonisation |
| IOD | Interocular difference |
| IRB | Institutional Review Board |
| ITT | Intention to treat |
| IXT | Intermittent exotropia |
| JCHR | Jaeb Center for Health Research |
| logMAR | Logarithm of the minimal angle of resolution |
| log sec arc | Logarithm of the seconds of arc |
| MCMC | Monte Carlo Markov chain |
| NIH | National Institutes of Health |
| Obs | Observation |
| PACT | Prism and alternate cover test |
| PEDIG | Pediatric Eye Disease Investigator Group |
| QA | Quality assurance |
| QC | Quality control |
| RBM | Risk-based monitoring |
| RCT | Randomized clinical trial |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SE | Spherical equivalent refractive error (Sphere + ½ Cylinder) |
| sec arc | Seconds of arc |
| SPCT | Simultaneous prism and cover test |
| VA | Visual acuity |

IXT7ProtV1.0\_19Apr2022 

#### PRINCIPAL INVESTIGATOR AGREEMENT FOR PROTOCOL

# Randomized Trial of Full-Time Occlusion Therapy for Intermittent Exotropia in Children (IXT7)

| Site | Numb | er: |
|------|----------|-----|
| | 1 (dillo | |

Each clinical site that is approved to participate in the IXT7 study will have one individual designated as the Protocol Principal Investigator (Protocol PI) at the site for that protocol. This may or may not be the same investigator that serves as the overall Site Principal Investigator (Site PI) for all PEDIG studies.

The Protocol PI and the Site PI (if different) agrees to the following for the IXT7 study. They will:

- Have a thorough understanding of the protocol design and study procedures.
- Ensure that local institutional requirements (if applicable) are satisfied for the protocol and that approvals and assurances are obtained annually if required.
- Ensure that the required protocol-certified staff, facilities, and equipment are available to conduct the protocol.
- Ensure that the required protocol staff have a thorough understanding of the protocol design and procedures.
- Provide adequate support and guidance to site investigators, coordinators, and other staff so that the study can be conducted according to protocol.
- Respond promptly to requests from the Coordinating Center (CC), Network Chair/s, or Protocol Chair/s.
- Correspond and maintain accessibility via email and phone with their PEDIG protocol monitor.
- Oversee local study documentation and records.
- Conduct periodic meetings of study personnel at their site.
- Cooperate with protocol monitors by working with the site coordinator to make available study personnel, study records, protocol binders, clinic charts for study participants, and other necessary records needed for on-site or virtual clinic monitoring visits.
- Notify the CC if any protocol adherence or data reporting problem is discovered or suspected.
- Attend scheduled PEDIG meetings and conference calls, including those for any PEDIG committees to which appointed.
- Review study monitoring reports evaluating clinical site performance and discuss with the CC any areas identified to be deficient.

The Protocol and PI shall exert diligent efforts to enroll at least three (3) study subjects.

In addition to the above, the Protocol PI and the Site PI (if different) agree(s) to the following:

- I/we understand the importance of successful follow-up of participants enrolled at my/our site.
- I/we agree as a site that we have the potential and commitment to as a site to enroll at least 3 subjects once certified.

| Protocol Principal Investigator's Signature | <b>Date:</b> // |
|---------------------------------------------|-----------------|
| Name: | |
| To be completed only if different: | |
| Site Principal Investigator's Signature | Date: / / |
| Name: | |

IXT7ProtV1.0 19Apr2022 

# PROTOCOL SUMMARY

| PARTICIPANT AREA | DESCRIPTION |
|---|---|
| Title | Randomized Trial of Full-Time Occlusion Therapy for Intermittent Exotropia in Children |
| Précis | Understanding the effectiveness of intensive patching has important implications for managing children with IXT. If full-time patching is associated with improvement in distance control vs an observation group, then future studies can be conducted to evaluate different durations of full-time patching treatment, whether the effect is maintained off-treatment, and how full-time patching compares to other treatment strategies. |
| Objectives | Determine whether full-time patching is more effective than observation for improving distance control of IXT after 3 months of treatment (ontreatment outcome). |
| Study Design | Randomized clinical trial. |
| Number of Sites | The study is open to all clinical sites approved to participate in the PEDIG network. |
| Endpoint | Primary Efficacy Outcome: Change in control of IXT at distance after 3 months based upon the average of three measures of control at distance. |
| | Key Safety Outcomes: |
| | 1. Deterioration is defined as meeting one of the following criteria at the 3 months follow-up visit: |
| | <ul> <li>Constant exotropia &gt;= 10∆ at distance AND near by SPCT. Constant is defined as an exotropia present throughout the examination and determined by at least three cover/uncover tests performed at various times during the exam. </li> <li>Decrease in near stereoacuity on the Randot Preschool Stereotest of at least 2 levels from baseline, or to nil.</li> </ul> |
| | 2. Decrease in distance visual acuity 3 or more logMAR lines from baseline in either eye or IOD 3 or more logMAR lines. |
| | 3. Diplopia 'More than 2 times per day' by parental report |
| | 4. Diplopia 'All the Time' by child symptom survey |
| Population | Inclusion Criteria: Children under the care of a pediatric optometrist or pediatric ophthalmologist will be eligible for the study if they meet all the following criteria: |
| | <ol> <li>Age 3 to &lt; 9 years</li> <li>IXT meeting all of the following criteria: <ul> <li>Intermittent or constant XT at distance (mean distance control 2.0 or more) with at least 1 control measure of 3, 4 or 5 (i.e., indicating spontaneous tropia)</li> <li>Either IXT, exophoria, or orthophoria at near (cannot have control score of 5 on all 3 near assessments)</li> <li>Distance exodeviation between 15Δ and 50Δ by PACT</li> <li>Near exodeviation between 0Δ and 50Δ by PACT</li> <li>Near exodeviation does not exceed distance by more than 10Δ by PACT (convergence insufficiency-type IXT excluded)</li> </ul> </li> <li>Age-normal visual acuity in both eyes: <ul> <li>3 years: 20/50 or better (&gt;=63 letters)</li> <li>4 years: 20/40 or better (&gt;=68 letters)</li> </ul> </li> </ol> |

IXT7ProtV1.0\_19Apr2022 

| PARTICIPANT AREA | DESCRIPTION |
|---|---|
| | <ul> <li>5-6 years: 20/32 or better (&gt;=73 letters)</li> <li>7-&lt;9 years: 20/25 or better (&gt;=78 letters)</li> <li>Interocular difference in distance VA of 2 logMAR lines or less (10 letters or less on E-ETDRS for patients ≥7 years old). Testing by ATS HOTV for participants 3 to &lt; 7 years old and by E-ETDRS for participants ≥7 years old.</li> <li>Cycloplegic refraction within the last 7 months.</li> <li>Refractive error between -6.00 D SE and +2.00 D SE (inclusive) based on a cycloplegic refraction within 7 months</li> <li>Participants with refractive error meeting any of the following based on a cycloplegic refraction within 6 months must be wearing spectacles for at least 2 weeks: <ul> <li>Myopia &gt; -0.50 D spherical equivalent (SE) in either eye</li> <li>Anisometropia &gt; 1.00 D SE</li> <li>Astigmatism in either eye &gt; 1.00 D</li> </ul> </li> <li>Any refractive correction worn at enrollment (required or not) must meet the following guidelines based on a cycloplegic refraction within 7 months: <ul> <li>Anisometropia SE must be within 0.50 D of the full anisometropic difference correction</li> <li>Astigmatism must be corrected within 0.50 D</li> <li>Axis must be within ±10 degrees if cylinder power is ≤1.00 D and within ±5 degrees if cylinder power is &gt;1.00 D.</li> <li>For hyperopia, the spherical component can be reduced at investigator discretion provided the reduction is symmetrical and does not meet the definition of deliberate overminus (see below).</li> <li>For myopia, the intent is to fully correct, but the spherical component can be undercorrected at investigator discretion provided the reduction is symmetrical and results in no more than -0.50 D SE residual (i.e., uncorrected) myopia. Deliberate overminus is not allowed.</li> <li>Deliberate overminus is defined for this protocol as any refractive correction prescribing reduced plus) is not consid</li></ul></li></ul> |
| | <ul> <li>For refractive errors with an emmetropic or myopic SE, the intent is to fully correct, but the spherical component can be undercorrected at investigator discretion provided the reduction is symmetrical and results in no more than -0.50 D SE residual (i.e., uncorrected) myopia. Prescribing a correction that yields more than 0.50 D <i>more minus</i> SE than the cycloplegic refraction SE is considered deliberate overminus and is not allowed.</li> <li>Note that the refractive correction guidelines and the requirement to wear refractive correction for at least 2 weeks apply not only to participants who require refractive correction under the above criteria but also to any other participant who is wearing refractive correction.</li> <li>Gestational age &gt; 30 weeks</li> <li>Birth weight &gt; 1500 grams</li> <li>Patient and/or parent understands protocol, is willing to enroll, and is willing to accept that other (i.e., nonrandomized) treatment for IXT will not be offered by the investigator for 3 months</li> <li>Parent has phone and is willing to be contacted by Jaeb Center staff</li> </ul> |

IXT7ProtV1.0\_19Apr2022 

| PARTICIPANT AREA | DESCRIPTION |
|---|---|
| | not anticipated |
| | Exclusion Criteria: |
| | Individuals meeting any of the following criteria at baseline will be excluded from study participation: |
| | <ol> <li>Prior strabismus, intraocular, or refractive surgery (including BOTOX injection)</li> <li>Prior nonsurgical treatment for IXT (e.g., patching, vergence therapy, vision therapy/orthoptics, base-in prism, or deliberate overminus (more than 1.00 D) spectacles of &gt;1 week duration within the past year</li> <li>Previous amblyopia treatment other than refractive correction</li> <li>Diplopia more than 2 times per day by parental assessment</li> <li>Paretic or restrictive strabismus</li> <li>Craniofacial malformations affecting the orbits</li> <li>Ocular disorders which would reduce VA (except refractive error)</li> <li>Severe developmental delay that would interfere with treatment or evaluation (in the opinion of the investigator). Participants with mild speech delay or reading and/or learning disabilities or ADHD are not excluded.</li> <li>Neurological anomaly that could affect ocular motility (e.g., cerebral palsy, Down syndrome)</li> <li>Immediate family member (child or sibling) of any investigative site personnel directly affiliated with this study.</li> </ol> |
| | 11. Known allergy to adhesive patches. 12. Known allergy to silicone. |
| Sample Size | 72 (36 observation, 36 full-time patching) |
| Phase | Phase 3 |
| Treatment Groups | Random assignment to: Observation Full-time patching (all waking hours, 7 days/week) |
| Participant Duration | 3 months after randomization |
| Protocol Overview/Synopsis | Participants will be randomly assigned to observation or full-time patching. All parents will receive a phone call at 4 weeks to answer any questions about observation or patching treatment. Participants will be followed for 3 months. |

IXT7ProtV1.0\_19Apr2022 

## STUDY SUMMARY FLOW CHART

#### Major Eligibility Criteria

- Children aged 3 to <9 years
- Intermittent exotropia meeting all the following criteria:
  Intermittent or constant XT at distance (mean distance control 2.0 or more, with at least 1 measure of 3, 4 or 5
  - IXT or exophoria or orthophoria at near (cannot have control score of 5 on all 3 near assessments)
  - Distance deviation between  $15\Delta$  and  $50\Delta$  by PACT
  - Near deviation between 0Δ and 50Δ by PACT
  - Near deviation does not exceed distance by more than 10Δ by PACT
- No prior strabismus, intraocular, or refractive surgery (including BOTOX injection)
- No previous nonsurgical treatment of >1 week duration within the past year
- No amblyopia treatment other than refractive correction
- No diplopia more than 2 times per day by parental report
- Refractive error between -6.00 D SE and +2.00 D SE (inclusive) based on a cycloplegic refraction within 7 months
- Age-normal VA (3 yrs = 20/50 or better; 4 yrs = 20/40 or better; 5-6 yrs = 20/32 or better; 7-8 yrs = 20/25 or better)
- No interocular VA difference more than 0.2 logMAR
- Wearing appropriate refractive correction for at least 2 weeks
- No abnormality of the cornea, lens, or central retina
- No known allergy to adhesive patches or silicone.

#### Enrollment/Baseline Visit

- · Informed consent
- Pediatric Eye Questionnaire (PedEyeQ)
- IXT Symptom Survey
- Diplopia Assessment by Parent
- Randot Preschool Stereoacuity (40 cm)
- Exotropia control #1 (distance and near)
- Divergence and convergence fusional amplitudes
- Exotropia control #2 (distance and near)
- Ocular alignment (cover/uncover, SPCT, PACT)
- Exotropia control #3 (distance and near)
- Suppression
- Retinal correspondence (ages 6-8 years)
- Assessment of eligibility



#### 3 months (±2 weeks) Primary Outcome

- Patch adherence monitoring (patching group only)
- Pediatric Eye Questionnaire (PedEyeQ)
- IXT Symptom Survey
- Diplopia Assessment by Parent
- Randot Preschool Stereoacuity (40 cm) (masked)
- Exotropia control #1 (distance and near) (masked)
- Divergence and convergence fusional amplitudes (masked)
- Exotropia control #2 (distance and near) (masked)
- Ocular alignment (cover/uncover, SPCT, PACT) (masked)
- Exotropia control #3 (distance and near) (masked)
- Suppression (masked)
- Retinal correspondence (ages 6-8 years) (masked)

 IXT7PROTV1.0 19Apr2022

# SCHEDULE OF STUDY VISITS AND PROCEDURES

| | Enrollment | 4-Week<br>Call | 3-Month<br>Visit |
|---|---|---|---|
| Consent | X | | |
| Demographics / Medical History | X | | |
| Treatment Compliance | | X | X |
| Quality of Life Survey | X | | X |
| IXT Symptom Survey | X | | X |
| Diplopia Assessment by Parent | X | | X |
| Distance Visual Acuity | X | | X |
| Randot Preschool Stereoacuity | X | | X |
| Exotropia Control (distance and near) | X | | X |
| Amplitude Testing (Divergence and Convergence) | X | | X |
| Ocular Alignment (distance and near) | X | | X |
| Suppression (distance) | X | | X |
| Retinal Correspondence* | X | | X |

<sup>&</sup>lt;sup>a</sup> Retinal correspondence to be measured only in children 6, 7, or 8 years of age at randomization

IXT7ProtV1.0\_19Apr2022 

# **Chapter 1: Background Information**

### 1.1 Epidemiology and Clinical Characteristics

- 3 Intermittent exotropia (IXT) is the most common form of childhood-onset exotropia, 1,2 with an
- 4 incidence of 32.1 per 100,000 in children under 19 years of age, and occurring more frequently
- 5 in females<sup>3</sup> and in Asian populations.<sup>4-6</sup> Onset of IXT is thought to be in the first year of life.<sup>7</sup>
- 6 Etiology is unknown although anatomical, innervational, sensory, and genetic factors have been
- 7 proposed.<sup>8,9</sup>

1

2

- 8 IXT is characterized by an exodeviation present predominantly at distance fixation with or
- 9 without deviation at near fixation. Pseudonyms include periodic exotropia and exotropia of
- inattention. In addition to being present for distance viewing, exotropia may also occur at near
- and with inattention, in bright sunlight, or when tired. Closure of one eye in bright sunlight and
- sensitivity to sunlight<sup>10-12</sup> are also characteristic features. Normal binocular single vision is
- typically present at near when the eyes are aligned, with normal (occasionally subnormal)
- stereoacuity. <sup>13,14</sup> Diplopia is rarely reported. <sup>15</sup>
- 15 IXT is characterized by unique sensory adaptations: 16 suppression mechanisms prevent diplopia
- when the exodeviation is manifest, but normal binocular single vision with normal stereoacuity is
- 17 reestablished when the deviation is controlled (albeit with persistent temporal retinal suppression
- in some children<sup>17</sup>). In addition, some children with IXT are thought to covary between normal
- and anomalous retinal correspondence (ARC)<sup>16,18</sup> and may also experience panoramic
- viewing.<sup>7,19</sup> However. the true nature of these adaptations, how often they occur, and how they
- 21 respond to treatment are poorly characterized having not been previously studied in large
- 22 numbers of children with IXT.

## 23 1.2 Current Management Strategies

- 24 IXT is currently managed by observation alone, or with surgical correction or non-surgical
- 25 treatment. 14 Despite a plethora of studies evaluating treatments for IXT, there are relatively few
- data on treatment effectiveness<sup>14</sup> and current practice patterns are fragmented.<sup>20,21</sup>
- 27 In addition, long-term success following treatment appears elusive, and specific reasons for
- 28 treatment failure are unclear. Popular explanations include the possibility that persistent sensory
- 29 maladaptations (suppression and/or anomalous retinal correspondence), as well as inadequate
- fusional amplitudes, may be responsible for recurrence of the exotropia following treatment.
- 31 To provide context for the proposed randomized clinical trial (RCT), the following summary
- briefly describes commonly used management strategies along with data from previous RCTs.

#### **1.2.1 Observation**

- 34 We are aware of two previous RCTs in which subjects with IXT were randomized to
- observation. The PEDIG IXT2 studies<sup>22,23</sup> randomized children to observation versus part-time
- patching. In the older cohort randomized to observation (3 to < 10 years at enrollment),
- deterioration of IXT (constant exotropia  $\ge 10\Delta$  at distance and near or  $\ge 2$ -octave decrease in near
- 38 stereoacuity from the best previous measure, or being prescribed treatment despite not having
- met motor or stereo deterioration) was met in 25 of 183 by 3 years (15%, 95% confidence
- interval = 10%-22%), 12 of whom were prescribed treatment without meeting motor or
- stereoacuity criteria.<sup>24</sup> However, of the 132 who completed the 3-year visit and had not been

- 42 treated during the study, only 1 (<1%) met motor or stereoacuity deterioration criteria at 3
- 43 years.<sup>24</sup> Of those older children randomized to observation who remained untreated over the 3
- years, "complete or near complete resolution" (exodeviation  $\leq 10\Delta$  at distance and near, no
- 45 reduction in stereoacuity, and no other nonsurgical treatment for IXT, having never met
- deterioration criteria) was met in 6 (7%) of 86.<sup>25</sup>
- 47 In the younger cohort randomized to observation (12-35 months at enrollment), deterioration of
- 48 IXT (constant exotropia ≥10 prism diopters at distance and near or treatment prescribed despite
- 49 not having met motor deterioration) occurred in 28% (95% CI = 20%–39%) by 3 years.<sup>26</sup> Of the
- 50 24 participants meeting the primary outcome of deterioration, seven met motor deterioration and
- 51 17 were prescribed treatment without meeting motor deterioration. <sup>26</sup> The cumulative probability
- of motor deterioration by 3 years was 10% (95% CI = 5%–19%).
- In a pilot RCT of surgery versus observation for IXT, Clarke et al<sup>27</sup> found 2 (9%) of 22 in the
- observation group showed significant improvement in control (improved 3 and 4 points on the
- office control scale) after 9 months of follow-up.

## 56 **1.2.2 Surgery**

- 57 The aim of surgery for IXT is to reduce the magnitude of the exodeviation (or eliminate it
- completely) such that any residual deviation can be easily compensated by existing convergence
- and divergence motor fusion mechanisms. Two RCTs have evaluated surgery for IXT. 14 PEDIG
- 60 (IXT1)<sup>28</sup> compared bilateral and unilateral surgery and found complete or near-complete
- resolution of IXT in 30% of participants overall at 3 years postoperatively (complete or near
- 62 complete resolution defined as exodeviation  $<10\Delta$  at distance and near, reduction of  $\ge10$   $\Delta$  by
- 63 PACT, esotropia  $<6\Delta$  by SPCT at distance and near, no >2 octave reduction in stereoacuity, no
- reoperation, no nonsurgical treatment for recurrent or residual exodeviation, and having never
- met failure criteria [exotropia  $> 10\Delta$  by SPCT at distance or near, constant esotropia  $> 6\Delta$  by
- SPCT at distance or near, and  $\geq 2$  octave reduction in stereoacuity]). In a separate RCT,
- Kushner<sup>29</sup> also compared unilateral versus bilateral surgery and found a satisfactory outcome
- (aligned within  $10\Delta$  of exophoria and  $5\Delta$  of esophoria) in 82% and 52% respectively, but
- outcomes were evaluated at only one year postoperatively. In IXT1, <sup>30</sup> younger age (3 to <5)
- years) was associated with a lower risk of failure by 3 years (28% vs 50%); however, reasons for
- failure versus success were not explored in Kushner's RCT.

## 72 1.2.3 Nonsurgical treatments

- 73 The aim of nonsurgical treatment for IXT is to improve the strength and/or quality of binocular
- single vision (reducing suppression, increasing fusional amplitudes), thereby improving control
- of the exodeviation. Commonly utilized non-surgical management strategies include, vision
- therapy, overminus lenses, relieving or correcting base-in prism, and part-time patching.

#### 77 Vision therapy:

- 78 There are no published RCTs of vision therapy, but a multicenter pilot RCT is planned and due
- 79 to commence in 2021 (NCT04487249).

## 80 Overminus optical correction:

- A recently published RCT (IXT5; NCT02807350) conducted by PEDIG,<sup>31</sup> randomized 3- to 10-
- years old with IXT to overminus spectacles (-2.50 D over cycloplegic refraction for 12 months)
- vs non-overminus spectacles and found better mean distance control at 12 months (in correction)

- 84 for participants treated with overminus spectacles (n=196) than those with non-overminus
- spectacles (n=190) (1.8 vs 2.8 points; adjusted difference, -0.8; 95% CI, -1.0 to -0.5; P < 0.001).
- 86 Factors associated with better versus worse control at outcome were not evaluated. However, a
- greater myopic shift occurred in those with overminus vs non-overminus treatment (-0.42 D vs
- 88 -0.04 D; adjusted difference, -0.37 D; 95% CI, -0.49 to -0.26 D; P<0.001), resulting in the
- 89 overminus spectacles being discontinued before follow-up was complete in some participants.<sup>31</sup>

## 90 **Prism correction:**

- 91 Relieving base-in prism correction was evaluated in an 8-week pilot RCT conducted by PEDIG
- 92 (IXT6; NCT03998670). The primary outcome was change in exodeviation control score, but
- 93 factors associated with success versus failure of treatment were not evaluated. Results are due to
- be published later this year.

## 95 **Patching:**

- Patching is one of the most frequently prescribed nonsurgical treatments for IXT and is described
- 97 in detail below (section 1.3).

98 99

100

## 1.3 Patching

## 1.3.1 Current clinical practice

- Prevailing clinical practice is to prescribe a low dose of 2-4 hours/day, and to either patch
- alternate eyes, alternate days, or patch the eye preferred for fixation (if present). Some clinicians
- prescribe for longer periods of time such as 6-8 hours/day or full-time (all waking hours) based
- on their clinical experience or outcomes from previous full-time patching studies, <sup>32,33</sup> but there is
- no evidence to support whether full-time patching has additional benefit to part-time patching.
- Patching may be prescribed over a short duration of weeks or months or may be utilized on and
- off over a period of years. It is currently prescribed either to improve exodeviation control to the
- point where other treatments are not necessary, or to maintain reasonable control until the child
- and family are ready for other treatments such as surgery or vision therapy. While patching
- therapy is thought to improve exodeviation control and potentially reduce the size of the
- exodeviation, there are few data on the magnitude of such effects or whether any benefit persists
- long-term.

#### 113 1.3.2 Previous Randomized Trials of Patching Treatment

- 114 Akbari et al 2020<sup>34</sup>: Akbari et al recently published a RCT<sup>34</sup> comparing part-time patching (2
- hours a day, alternating eyes) to observation in 76 children who were 3- to 8-years-old with IXT.
- The primary outcome was a single measure of control, using a modification of the Office Control
- Score<sup>35</sup> at 3 and 6 months (on treatment). Control scores ranged from 0 (phoria) to 6 (constant
- exotropia) and were better (lower score) in the patching group at 3 months (distance: 2.3±1.0
- points vs 2.7 $\pm$ 1.1 points; P=0.03; near: 1.2 $\pm$ 0.7 points vs 1.5 $\pm$ 0.6 points; P=0.003), and at 6
- months (distance:  $2.4\pm1.1$  points vs  $2.8\pm1.2$  points; P=0.03; near:  $1.0\pm0.6$  points vs  $1.6\pm0.9$
- points; P=0.003). Nevertheless, post-treatment outcomes, as well as effects on suppression, angle
- of deviation, and fusional amplitudes were not evaluated. In addition, while control improved
- with patching, control scores reflect that many participants had persistent intermittent exotropia.
- PEDIG 2014<sup>22</sup> and PEDIG 2015<sup>23</sup>: Two PEDIG RCTs evaluated part-time patching (3 hours a
- day for 5 months) versus observation in 12- to 35-month-olds<sup>23</sup> and 3- to <11-year-olds<sup>22</sup> with
- 126 IXT. In published secondary analyses of 6-month outcomes (1-month post cessation of patching

IXT7ProtV1.0 19Apr2022 

- treatment), mean control scores and mean angle of deviation were compared between patching
- and observation groups. For 12- to 35-month-olds, mean distance control scores were better
- (lower) in the patching group compared with the observation group (2.3 points vs 2.8 points;
- 130 P=0.02) (near control scores were similar: 1.1 points vs 1.4 points; P=0.26).<sup>23</sup> In addition, mean
- distance angle of deviation (PACT) was significantly smaller in the patched group (24.9 $\Delta$  vs
- 132 27.9Δ, P=0.02)(near angle was similar: 17.0Δ vs 19.3Δ, P=0.10). For 3- to <11-year-olds,
- distance control scores were similar between groups (2.0 points patching vs 2.3 points
- observation; P=0.094) but near control scores were lower in the patching group (0.9 points vs 1.2
- points; P=0.013). Mean angle of deviation by PACT was 22.2 $\Delta$  in the patching group vs 23.8 $\Delta$
- in the observation group (P=0.012) at distance and 15.4 $\Delta$  vs 17.6 $\Delta$  (P=0.11) at near.
- 137 The studies were designed primarily to evaluate deterioration rates, but in post hoc analyses
- 138 (publication in process) of 3- to <11-year-olds with a control score of 2 or more at enrollment
- and a 3-month on-treatment examination (matching current study inclusion criteria and primary
- outcome time-point) distance control improved 0.4 points in the observation group (n=147) and
- 0.8 points in the patching group (n=125) (mean difference 0.41 points (95% CI, 0.12 to 0.70)
- points). Angle of deviation improved  $0.2\Delta$  in the observation group and  $2.3\Delta$  in the patching
- group (mean difference  $2.1\Delta$  (0.6 to 3.6 $\Delta$ ).
- Nevertheless, in both the 12- to 35-month and 3- to <11-year-old cohorts, many participants had
- persistent intermittent exotropia post-treatment. Changes in suppression or fusional amplitudes,
- and relationships with better versus worse control, were not evaluated.

## 1.3.3 Previous Non-randomized Studies of Patching Treatment

- A small number of non-randomized studies have evaluated patching for IXT. 16,36,37 While there
- are intrinsic challenges when interpreting data from non-randomized studies, the following are
- selected for more detailed review either because they provide additional information on potential
- effects of full-time patching, and/or provide some insight regarding how patching may impact
- sensory adaptations, the angle of deviation, or fusional amplitudes.

## 153 Full-time Patching

- 154 Iacobucci & Henderson 1965<sup>33</sup>: Twenty-eight children with IXT, scheduled for surgery, were
- selected ("at random") for full-time patching for 3 months. IXT control and angle of deviation
- were compared with a control group of 38 children undergoing anti-suppression and diplopia
- therapy. Distance angle of deviation by PACT reduced by a mean of  $5.8\pm1.1\Delta$  from baseline to 3
- months in the patching group, compared with an increase of  $1.8\pm0.4\Delta$  in the control group. Near
- angle of deviation by PACT reduced by a mean of  $4.6\pm1\Delta$  from baseline to 3 months in the
- patching group, compared with an increase of  $1.3\pm0.5\Delta$  in the control group. Eleven of 28
- patched patients and 20 of 38 control patients were constant exotropia at distance at baseline; of
- these, 8 (73%) of 11 in the patching group and 0 of 20 in the control group became intermittent
- or phoric at 3 months.
- 164 <u>Flynn et al 1976<sup>32</sup>:</u> In a prospective study, Flynn and colleagues prescribed full-time patching for
- 4-12 weeks to 31 children (mean age 7.6 years, range 3 to 13 years) with IXT. Mean angle of
- deviation pre-treatment was  $20\pm7\Delta$  at distance and  $15\pm12\Delta$  at near. Nine of 31 had undergone
- previous surgery. Following patching treatment, 7 (23%) of 31 showed dramatic improvement
- such that "the deviation became almost completely phoric, fusion improved, and all evidence of
- suppression on the synoptophore or in free space disappeared." Fourteen of 31 patients had a
- 170 reduction in angle of deviation and a change from tropia to intermittent tropia or phoria. In 12 of

- 171 31 patients there was a measurable improvement in suppression with disappearance of the
- suppression scotoma. Increase in the range of fusional amplitudes occurred in 9 of these 12
- patients. Of note, Flynn et al<sup>32</sup> report that some patients did not respond positively to patching,
- with 12 showing an increase in angle of deviation (mean  $5\Delta$ , range  $2\Delta$  to  $15\Delta$ ) and 6 showing
- worsening control. Long-term follow-up was not reported.

## 1.4 Mechanism of Patching Treatment Effect

- 177 Patching is considered "anti-suppression" therapy, affecting exodeviation control by reducing or
- eliminating the suppression that occurs when the exodeviation is manifest. 32,33,38,39

## **1.4.1 Suppression**

- Previous studies have attempted to evaluate the presence versus absence of suppression, as well
- as the size and location of the suppression scotoma when the exodeviation is manifest, <sup>15,18,40-44</sup>
- but few have evaluated changes in suppression with treatment or the relationship between
- suppression status and treatment success. In fact, although patching is designated "anti-
- suppression" treatment, there are few data demonstrating that changes in suppression occur with
- patching.

176

- 186 It has been suggested that, left untreated, suppression in many children with IXT will increase, 41
- making it harder to remediate and leading to poorer treatment outcomes, but this has not been
- studied. It has also been suggested that eradication of suppression is required for successful
- treatment, 15 but this deserves further study.

## 190 1.4.2 Fusional Vergence Amplitudes

- 191 Motor fusion mechanisms are responsible for maintaining binocular alignment, and in IXT, both
- 192 convergence and divergence are thought to be important for enabling motor control of the
- exodeviation. 45,46 In previous studies, 32,38,47,48 data suggest that patching results in an increase in
- 194 convergence amplitudes, but further study is needed to verify whether such changes truly occur
- and if they do, whether they are directly related to changes in suppression or occur
- independently. It is also unknown how such changes relate to improvement or successful
- treatment of IXT.

## 198 1.4.3 Magnitude of Deviation

- Previous studies<sup>22,23,32,33,39,48-50</sup> have shown that the magnitude of the deviation may reduce with
- 200 patching treatment. Nevertheless, there are few data that support this notion, and the mechanism
- by which patching might alter ocular alignment remains unclear.

## 202 1.5 Measuring Patch Wear Time

- Adherence with a prescribed patching dose is often problematic and limits the interpretation of
- findings when attempting to correlate dose to outcome. In studies of patching treatment for
- amblyopia, some research groups have used occlusion dose monitors (ODMs) to record actual
- 206 patch wear time. 51-54 In general these previous studies concluded that dose is a significant factor
- in determining amblyopia treatment outcome, although there remains considerable individual
- variability. We are unaware of previous studies that have analyzed actual patch wear time when
- treating IXT, and such data are important for understanding whether there is a dose effect
- 210 relationship.
- Recently, a new method of monitoring patching adherence has become available and is being
- used in a concurrent PEDIG amblyopia study (ATS22, NCT04378790). TheraMon®, a

| 213<br>214<br>215<br>216<br>217<br>218<br>219<br>220 | thermosensor device, appears to work well for monitoring adherence with amblyopia patching treatments in children. <sup>51</sup> We propose utilizing the TheraMon® in the current study to enable important secondary analyses of outcome in relation to actual (rather than prescribed) wear time. |
|---|---|
| | <b>1.6 Unanswered Questions Regarding Patching Treatment for IXT</b> While previous data confirm an effect of patching on control of IXT, and even on angle of deviation, there remain many unanswered questions regarding treatment effectiveness. Such questions include: |
| 221<br>222 | - Is prescribed full-time patching more effective for improving control and/or reducing angle of deviation than observation alone? |
| 223<br>224<br>225 | <ul> <li>Does patching alter suppression, angle of deviation, fusional amplitudes, or<br/>anomalous retinal correspondence, and are such changes related to exodeviation<br/>control?</li> </ul> |
| 226<br>227 | - Is there a dose-response relationship (greater improvement with more actual patching time)? |
| 228<br>229 | <ul> <li>Which clinical and demographic characteristics, if any, are associated with<br/>improvement in exodeviation control and/or treatment success?</li> </ul> |
| 230<br>231<br>232<br>233<br>234<br>235<br>236 | 1.7 Rationale for Present Study IXT is a common eye condition, but long-term surgical treatment outcomes are disappointing, with high failure rates due to recurrence or undercorrection of the exodeviation. Patching is a commonly used nonsurgical treatment for which there is some evidence of short-term treatment benefit (improved exodeviation control and reduced angle of deviation) when prescribed 2-3 hours/day. Nevertheless, the extent to which patching is effective if worn for long periods of time per day or if any treatment effect is sustained once treatment is discontinued is unknown. |
| 237<br>238<br>239<br>240<br>241<br>242 | Understanding the effectiveness of patching treatment and whether there is a benefit from full-time patching versus observation alone has important implications for managing children with IXT. If full-time patching is associated with more improvement in distance control compared to observation alone, then future studies can be conducted to evaluate different durations of full-time patching treatment, whether the effect is maintained off-treatment, and how full-time patching compares to other treatment strategies. |
| 243<br>244<br>245<br>246<br>247 | In addition, this study would provide evidence of the ability of patching to alter suppression, anomalous retinal correspondence, and fusional amplitudes, and the relationships of these clinical characteristics with treatment success, failure, and improvement of IXT. This study provides an opportunity to explore such relationships, and data are expected to create hypotheses for future studies. |
| 248 | 1.8 Study Objectives |
| <ul><li>249</li><li>250</li></ul> | Determine whether full-time patching is more effective than observation for improving distance control of IXT after 3 months of treatment (on-treatment outcome). |

 IXT7ProtV1.0\_19Apr2022

250 251

### 1.9 Potential Risks and Benefits of Study Treatment

#### 253 1.9.1 Known Potential Risks

- 254 There is a risk that patching may create diplopia that then becomes troublesome to the patient,
- but this complication is seldom reported. It is possible that some patients will show worsening of
- 256 IXT control or increase in magnitude with patching<sup>32</sup> or observation,<sup>22</sup> but deterioration criteria
- will be assessed after 3 months and the short 3-month duration allows for cessation of patching
- 258 treatment and/or commencement of other treatment should deterioration of the IXT occur. Skin
- 259 irritation may occur. If persistent skin irritation occurs due to the adhesive patch, the participant
- will be provided with a fabric patch to wear on their glasses (plano glasses will be provided for
- 261 children who are not already wearing glasses). Patching could potentially cause a decrease of VA
- in the patched eye, but that is very unlikely since alternating patching is prescribed, and any
- 263 decrease in VA is almost always reversible. One potential risk with observing IXT without
- 264 treatment is that suppression may increase in density over time. An increase in the density of
- suppression may predispose the child to worse motor and sensory outcomes in the long term, but
- with a 3-month study duration there is unlikely to be a significant change, and furthermore this
- has not been previously studied to know if and when this occurs.

#### 268 1.9.2 Known Potential Benefits

- The potential benefits of patching are improved exodeviation control, reduced angle of deviation,
- 270 reduced suppression, and/or increased fusional amplitudes.
- There are no direct benefits of observation, however, in a previous RCT, approximately 7% of
- 272 patients<sup>55</sup> resolved spontaneously over 3 years. Therefore, avoiding the need for treatment of
- 273 IXT and any associated risks of IXT treatment may be considered an indirect benefit of
- observation.

#### 275 1.10 Risks of Examination or Testing Procedures

- The procedures in this study are part of daily eye care practice in the United States and pose no
- known risks. As part of a routine usual-care exam, the participant may receive
- 278 cycloplegic/dilating eye drops.

279280

252

#### 1.11 Risk Assessment

- There are no risks involved in this study that would not be part of usual care when treating with
- 282 either patching or by observation alone. The protocol's level of risk is consistent with 45 CFR
- 283 46.404 and 21 CFR 50.51, which indicates research not involving greater than minimal risk for
- the individual child involved in the research.

285 286

#### 1.12 General Considerations

- The study is being conducted in compliance with the policies described in the PEDIG network
- 288 policies document, with the ethical principles that have their origin in the Declaration of
- Helsinki, with the protocol described herein, and with the standards of Good Clinical Practice
- 290 (GCP).

IXT7ProtV1.0 19Apr2022 

## **Chapter 2: Study Enrollment and Randomization**

## 2.1 Participant Recruitment and Enrollment

The study plans to enroll enough participants, for whom informed consent will be obtained, in order to randomize a minimum of 72 participants.

As the randomization goal approaches attainment, sites will be notified of the end date for recruitment into the study. Participants who have signed informed consent forms are enrolled and can be randomized until the end date, which means the expected recruitment number might be exceeded. The maximum number randomized will be 82

There is no restriction on the number of participants to be enrolled by each site toward the overall recruitment goal. The overall number of participants with an interocular difference in distance VA of 2 logMAR lines (10 letters on E-ETDRS for patients ≥7 years old) will be limited to 14.

#### 2.1.1 Informed Consent

Children with IXT who are 3 to <9 years of age attending ophthalmology or optometry outpatient visits will be identified.

Families who qualify for the study will be approached by one of the research team members. The study will be discussed with the child's parent(s) or guardian(s) [referred to subsequently as parent(s)]. Parent(s) who express an interest in the study will be given a copy of the informed consent form to read. Written informed consent must be obtained from a parent and written or verbal assent from the child (depending on age and local IRB requirements) prior to performing any study-specific procedures that are not part of the child's routine care.

A child is considered enrolled into the study when the informed consent form has been signed by the parent, the assent form has been signed by the child (when applicable), and the investigator has also signed the appropriate forms.

## 2.2 Eligibility Criteria

#### 2.2.1 Inclusion Criteria

Children under the care of a pediatric optometrist or pediatric ophthalmologist, who are identified during a standard-of-care outpatient visit or from a referral from another provider, will be eligible for the study if they meet all the following criteria:

- 1. Age 3 to  $\leq$  9 years
- 2. IXT meeting all the following criteria:
  - Intermittent or constant XT at distance (mean distance control 2.0 or more) with at least 1 measure of 3, 4 or 5 (i.e., indicating spontaneous tropia) on control testing
  - Either IXT, exophoria, or orthophoria at near (cannot have control score of 5 on all 3 near assessments)
  - Distance exodeviation between  $15\Delta$  and  $50\Delta$  by PACT
  - Near exodeviation between  $0\Delta$  and  $50\Delta$  by PACT
  - Near exodeviation does not exceed distance by more than 10Δ by PACT
- 3. Age-normal visual acuity in both eyes: 56-58


- 3 years: 20/50 or better (>=63 letters)
- 4 years: 20/40 or better (>=68 letters)

338

339

340341

342

343

344

345

346

347

348

349350

351

352

353

354

355

356357

358

359

360361

362

363

364365

366

367

368369

370

371372

373

374375

376

377378

379

380

381

- 5-6 years: 20/32 or better (>=73 letters)
- 7-<9 years: 20/25 or better (>=78 letters)
- 4. Interocular difference in distance VA of 2 logMAR lines or less (10 letters or less on E-ETDRS for patients ≥7 years old). Testing by ATS HOTV for participants 3 to < 7 years old and by E-ETDRS for participants ≥7 years old.
  - The overall number of participants with an interocular difference in distance VA of 2 logMAR lines (10 letters on E-ETDRS for patients ≥7 years old) will be limited to 14.
- 5. Refractive error between -6.00 D SE and +2.00 D SE (inclusive) based on cycloplegic refraction performed within 7 months
- 6. Participants with refractive error meeting any of the following based on cycloplegic refraction performed within the prior 7 months must be wearing spectacles for at least 2 weeks:
  - Myopia > -0.50 D spherical equivalent (SE) in either eye
  - Anisometropia > 1.00 D SE
  - Astigmatism in either eye > 1.00 D
- 7. Any refractive correction worn at enrollment (required or not) must meet the following guidelines based on cycloplegic refraction performed within the prior 7 months:
  - Anisometropia SE must be within 0.50 D of the full anisometropic difference correction
  - Astigmatism must be corrected within 0.50 D
  - Axis must be within  $\pm 10$  degrees if cylinder power is  $\leq 1.00$  D and within  $\pm 5$  degrees if cylinder power is  $\geq 1.00$  D.
  - For hyperopia, the spherical component can be reduced at investigator discretion provided the reduction is symmetrical and does not meet the definition of deliberate overminus (see below).
  - For refractive errors with an emmetropic or myopic SE, the intent is to fully correct, but the spherical component can be undercorrected at investigator discretion provided the reduction is symmetrical and results in no more than -0.50 D SE residual (i.e., uncorrected) myopia. Deliberate overminus is not allowed.
  - Deliberate overminus is defined for this protocol as any refractive correction prescribed to yield lenses that are overminused by more than -0.50D SE than cycloplegic refraction SE.
    - Less than the full cycloplegic hyperopic correction (i.e., prescribing reduced plus) or no correction for a hyperopic SE refractive error is not considered the same as overminusing for this protocol (because most patients without IXT but with hyperopic SE refractions up to +2.00 D SE would not typically be prescribed a refractive correction.)
  - Note that the refractive correction guidelines and the requirement to wear refractive correction for at least 2 weeks apply not only to participants who require refractive correction under the above criteria but also to any other participant who is wearing refractive correction.
- 8. Gestational age > 30 weeks

IXT7ProtV1.0 19Apr2022 

- 382 9. Birth weight > 1500 grams
- 383 10. Patient and/or parent understands protocol, is willing to enroll, and is willing to accept that other treatment for IXT will not be offered for 3 months
  - 11. Parent has phone and is willing to be contacted by Jaeb Center staff
  - 12. Relocation outside of area of an active PEDIG site within next 3 months not anticipated

## 387 388 389

390

391

392

393

394

395

396

397

398 399

400

401

402 403

404

405

406

407

385

386

#### 2.2.2 Exclusion Criteria

Individuals meeting any of the following criteria at baseline will be excluded from study participation.

- 1. Prior strabismus, intraocular, or refractive surgery (including BOTOX injection)
- 2. Prior nonsurgical treatment for IXT (e.g., patching, vergence therapy, vision therapy/orthoptics, base-in prism, or deliberate overminus with spectacles more than 1.00 D) for >1 week duration within the past 1 year
- 3. Previous amblyopia treatment other than refractive correction
- 4. Diplopia more than 2 times per day by parental assessment
- 5. Paretic or restrictive strabismus
- 6. Craniofacial malformations affecting the orbits
- 7. Ocular disorders which would reduce VA (except refractive error)
- 8. Severe developmental delay that would interfere with treatment or evaluation (in the opinion of the investigator). Participants with mild speech delay or reading and/or learning disabilities or ADHD are not excluded.
- 9. Neurological anomaly that could affect ocular motility (e.g., cerebral palsy, Down syndrome)
- 10. Immediate family member (child or sibling) of any investigative site personnel directly affiliated with this study.
- 11. Known allergy to adhesive patches.
- 12. Known allergy to silicone.

## 408 409 410

#### 2.3 Historical Information

Historical information elicited will include the following: date of birth, sex, race, ethnicity, spectacle correction, and prior treatment for IXT and amblyopia.

## 413 414

419

420

421

423

424

## 2.4 Screening and Baseline Procedures

- Testing will be done in the order specified below on a single day following enrollment in the
- 416 child's current refractive correction if worn (any spectacle correction worn must meet the criteria
- specified in section 2.2) and without cycloplegia:
- 1. Eye-Related Quality of life: Pediatric Eye Questionnaire (PedEyeQ)
  - Child questionnaire: Completed by children 5 years and older
  - Parent questionnaire: Completed by the parent for all children regardless of age (includes parent and proxy questions)

## 422 2. <u>Symptom Survey</u>:

- Intermittent Exotropia Symptom Survey completed by children 5 years or older.
- Single diplopia question to be completed by children 3 or 4 years.

IXT7ProtV1.0 19Apr2022 

- 3. <u>Diplopia Assessment by Parent</u>: Assess diplopia presence and frequency over the last week, by parental report. If present, classify diplopia frequency as "2 times or less per day" or "more than 2 times per day."
- 428 4. Monocular Distance VA Testing: Distance VA testing will be performed by a certified examiner on a certified VA system (EVA or M&S), using the ATS single surround HOTV for participants 3 to <7 years old and using the E-ETDRS for participants ≥ 7 years. The same VA testing method used at enrollment will be used again at 3 months.</li>
- 5. <u>Stereoacuity Testing:</u> Assessed using the Randot Preschool Stereotest at near (performed at 40 cm) as outlined the *IXT7 Procedures Manual*
- 6. Control of the Exodeviation #1: Control of the exodeviation at distance (6 meters) then near (1/3 meter) will be assessed using the standardized IXT control scale, 35 as outlined in the *IXT7 Procedures Manual*.
  - Testing must be performed by a pediatric ophthalmologist, pediatric optometrist, or certified orthoptist.
  - The same examiner must assess control for all three assessments of control at each visit.
  - 8. <u>Divergence Amplitude Testing</u>: Measured at distance (6 meters) using the PEDIG-approved prism bar as described in the *IXT7 Procedures Manual* 
    - Testing must be performed by a pediatric ophthalmologist, pediatric optometrist, or certified orthoptist.
    - Record the break and recovery points.
  - 9. <u>Convergence Amplitude Testing:</u> Measured at distance (6 meters) using the PEDIG-approved prism bar as described in the *IXT7 Procedures Manual* 
    - Testing must be performed by a pediatric ophthalmologist, pediatric optometrist, or certified orthoptist.
  - 10. Control of the Exodeviation #2 (repeat) (see item #7).
  - 11. Ocular Alignment Testing:

437 438

439

440

441

442

443 444

445

446

447 448

449

450

451

452

453

454 455

456

457

458

459

460

461

462

463

464 465

466

467

- Testing must be performed by a pediatric ophthalmologist, pediatric optometrist, or certified orthoptist.
- Ocular alignment will be assessed by the cover/uncover test, simultaneous prism and cover test (SPCT), and prism and alternate cover test (PACT) in primary gaze at distance (3 meters) and near (1/3 meter) as described in the *IXT7 Procedures Manual*.
- 12. Control of the Exodeviation #3 (repeat) (see item #7)
- 13. <u>Suppression:</u> Assessment of suppression at distance (6 meters) using the Office Suppression Test<sup>59</sup> as described in the *IXT7 Procedures Manual* 
  - Testing must be performed by a pediatric ophthalmologist, pediatric optometrist, or certified orthoptist.
- 14. <u>Retinal Correspondence (children 6 to <9 years only):</u> Assessment of retinal correspondence will be made when aligned and also when tropic using the Hering-Bielschowsky After Image Test<sup>60</sup> as described in *the IXT7 Procedures Manual* using the PEDIG-supplied flash unit.
  - Testing must be performed by a pediatric ophthalmologist, pediatric optometrist, or certified orthoptist.

IXT7ProtV1.0 19Apr2022 

#### 2.5 Randomization

- Eligible participants will be randomly assigned on the study website to the following treatment:
- 470 471

468

- 1. Observation for 3 months no treatment other than refractive correction
- 472 2. Full-time patching (all waking hours) for 3 months (right eye on even days, left eye on odd days), in addition to refractive correction

474

491

492

- The Jaeb Center will construct a Master Randomization List stratified by mean distance control
- score at enrollment (2 to <3, 3 to <4, 4 to 5). A participant is officially randomized when the
- website randomization process is completed.

## 478 **2.5.1 Observation Group**

- 479 Participants randomized to observation alone will not be allowed to receive any other treatment
- 480 for IXT, except refractive correction, for 3 months.

## 481 **2.5.2 Full-Time Patching Group**

- Participants randomized to the full-time patching group will patch full-time (all waking hours)
- for 3 months up until the day before the 3-month primary outcome visit. Daily alternate patching
- will be prescribed (right eye on even days, left eye on odd days). No other treatment for IXT will
- be used, except for refractive correction.

## 486 **2.6 Monitoring of Adherence**

- 487 Site staff will activate and distribute occlusion dose monitors (ODMs) for participants
- randomized to patching (patching adherence is not applicable to the observation group).
- Adherence with patching will be monitored throughout the study by an ODM worn on the inside of the patch for participants randomized to patching.
  - In addition, parents will be asked to record patching wear time and which eye was patched on a study calendar.

IXT7ProtV1.0 19Apr2022 

#### **Chapter 3: Study Follow-up** 493 494 3.1 Study Visits 495 Study follow up for participants randomized in the study is (timed from randomization): 496 497 • 4-week phone call: 4 weeks $\pm$ 1 week 498 • 3-month (on treatment) primary outcome visit: 3 months $\pm$ 2 weeks 499 • Parents will be instructed to not patch on the day of the visit 500 3.2 Phone Call at 4-weeks 501 502 Study personnel will call the parent of each participant 4 weeks $\pm$ 1 week following 503 randomization. The purpose of the call for the patching groups is to determine whether patching 504 is being done, and if so, how it is being done. If patching is not being done correctly, patching 505 instructions will be reviewed with the parents. Parents in the patching groups will be asked if 506 they have had any problems using the ODM. If ODMs have been lost, replacement ODMs may 507 be sent to the parent. Parents in both treatment groups will be asked if they have any questions or 508 concerns about the study. 509 3.3 Masking Procedures 510 Participants will not be masked to their treatment group, given that they will be asked to patch all 511 waking hours/day (full-time patching group) or not at all (observation group). The investigator treating each participant also will not be masked to treatment group. An examiner masked to 512 513 treatment group will perform all clinical testing (with the exception of VA testing and 514 administration of questionnaires, which may be performed by unmasked, certified personnel) at 515 the 3-month visit. 516 3.3.1 Masked Examiner 517 The masked examiner must be a pediatric optometrist, pediatric ophthalmologist, or certified 518 orthoptist who is not aware of the participant's assigned treatment. Because the enrolling 519 investigator will be unmasked to treatment group, they will not be allowed to serve as their own 520 masked examiner. 521 3.4 Testing Procedures at 3-Month Outcome Visit 522 The following procedures will be performed in the order specified below at the 3-month outcome 523 visit with the participant wearing their current refractive correction (if worn), and without 524 cycloplegia. If unable to complete the entire masked exam during the office visit, the participant 525 can return with 10 days to complete all masked testing (#6-14 below). Testing procedures #1-5 526 below do not need to be repeated if completed at the initial office visit. 527 528 1. Adherence Monitoring (for patching group): • Evaluate compliance by review of study calendar 529 530 • Download adherence data from ODM 531 2. Eye-Related Quality of life: Pediatric Eye Questionnaire (PedEyeQ) 532 • Child questionnaire: Completed by children 5 years and older 533 • Parent questionnaire: Completed by the parent for all children regardless of age 534 (includes parent and proxy questions) 535 3. Symptom Survey:

IXT7ProtV1.0 19Apr2022 

- Intermittent Exotropia Symptom Survey completed by children 5 years or older.
- Single diplopia question to be completed by children 3 or 4 years.
- 538 4. <u>Diplopia Assessment by Parent</u>: Assess diplopia presence and frequency over the last week, 539 by parental report. If present, classify diplopia frequency as "2 times or less per day" or 540 "more than 2 times per day."
- 541 5. Monocular Distance VA Testing: Distance VA testing in each eye using the same test method used at enrollment.
- 6. <u>Stereoacuity Testing (masked)</u>: Randot Preschool Stereoacuity at 40 cm.
- 7. Control of the Exodeviation #1 (masked):
  - Distance (6 meters)
  - Near (1/3 meter)

545

546

547

548

549

550

553

555

556557

558559

560

561

562563

564

565

566567

568569

- The same examiner must assess control for all three assessments of control for each visit.
- 8. <u>Divergence Amplitude Testing (masked)</u>: Measured at distance (6 meters) using a PEDIG-approved prism bar as described in the *IXT7 Procedures Manual* 
  - Record the break and recovery points
- 9. <u>Convergence Amplitude Testing (masked)</u>: Measured at distance (6 meters) using a PEDIGapproved prism bar as described in the *IXT7 Procedures Manual* 
  - Record the blur, break, and recovery points
- 10. <u>Control of the Exodeviation #2 (masked)</u> (repeat) (see item #7)
  - 11. Ocular Alignment Testing (masked):
    - Testing must be performed by a pediatric ophthalmologist, pediatric optometrist, or certified orthoptist.
    - Ocular alignment will be assessed by the cover/uncover test, simultaneous prism and cover test (SPCT), and prism and alternate cover test (PACT) in primary gaze at distance (3 meters) and near (1/3 meter) as described in the *IXT7 Procedures Manual*.
  - 12. Control of the Exodeviation #3 (masked) (repeat) (see item #7)
  - 13. <u>Suppression (masked)</u>: Assessment at distance using the Office Suppression Test at distance (6 meters) as described in the *IXT7 Procedures Manual*
  - 14. <u>Retinal correspondence (masked)</u>: In children aged 6, 7, or 8 years of age at randomization, assessment of retinal correspondence will be made using the Hering-Bielschowsky After-Image Test as described in *the IXT7 Procedures Manual* using the PEDIG-supplied flash unit.

## 3.5 IXT Treatment Changes During Follow-up

- 570 Changes in treatment are not allowed prior to the 3-month outcome visit.
- 571 If the participant is experiencing overwhelming social concerns or significant symptoms
- associated specifically with IXT, the investigator <u>must call one of the Protocol Chairs</u> to
- discuss the case and obtain approval for an early 3-month outcome visit (if not already in
- window) prior to initiating any non-randomized treatment for IXT.
- 575 3.6 Management of Refractive Error During Follow-up
- Because of the short duration of the study, the spectacles prescribed at randomization may not be
- 577 changed or discontinued without contacting a Protocol Chair.

IXT7ProtV1.0 19Apr2022 

- In the event that spectacles are lost or damaged after randomization but before the 3-month outcome visit, the spectacles may only be replaced with the same spectacle prescription that was
- prescribed at randomization.

IXT7ProtV1.0\_19Apr2022 

## **Chapter 4: Testing Procedures and Questionnaires**

#### 582 4.1 Clinical Assessments

581

- The following test procedures will be completed for all three treatment groups at each visit as defined in the *IXT Procedures Manual*:
- Monocular VA Testing: Distance VA will be tested in both eyes with the participant wearing their study-specified spectacle correction. The right eye is tested, with the left eye occluded with an adhesive patch. The left eye is tested after the right eye. Testing must be performed by a certified examiner on a certified VA system (EVA or M&S), using the ATS single surround HOTV for participants 3 to <7 years old and using the E-ETDRS for participants ≥ 7 years. The same testing method must be used throughout the study. Testing time for both eyes typically is in the range of 5 to 10 minutes.</li>
- 592 2. Randot Preschool Stereoacuity Test: The Randot Preschool Stereoacuity Test measures 6 593 levels (40 to 800 seconds of arc) of stereoacuity at near (40 cm). The test consists of 3 594 booklets, each designed to test 2 levels of stereoacuity, and each level consisting of 4 panels, 595 3 of which contain a random dot stereogram. The participant wears polarized lenses over 596 their spectacle correction. The examiner asks the participant if they can identify a specific 597 black and white shape in the booklet and then asks the participant to point to the panel 598 containing the corresponding stereogram image, as outlined in the IXT7 Procedures Manual. 599 The test must be administered by a certified examiner. The certified examiner will be 600 required to be masked to treatment group. Testing time is approximately 2-4 minutes.
- 3. Ocular Alignment: Ocular alignment will be assessed by the cover/uncover test, simultaneous prism and cover test when tropia present by cover/uncover test (SPCT), and prism and alternate cover test (PACT), using the PEDIG-approved IXT7 prism bar, in primary gaze at distance (6 meters) and at near (33 cm) as outlined in the *IXT7 Procedures Manual*. The examiner will be required to be masked to treatment group. Testing time is approximately 2-4 minutes.
- 607 4. <u>Cycloplegic Refraction</u>: A cycloplegic refraction will be done prior to enrollment and only if
   608 clinically indicated thereafter. After administration of eye drops, it typically takes 30 minutes
   609 to achieve cycloplegia, and testing time for refraction of both eyes is in the range of 2 to 10
   610 minutes.
- 5. <u>Suppression Testing:</u> Suppression will be assessed using the Office Suppression Test which grades the level of suppression while tropic on a 4-level scale. Testing will be performed at 6 meters as outlined in the *IXT7 Procedures Manual*. Testing must be performed by a pediatric ophthalmologist, pediatric optometrist, or certified orthoptist. The examiner will be required to be masked to treatment group. Testing time is approximately 3-5 minutes.
- 6. Retinal Correspondence Testing: In children 6, 7, or 8 years old at time of randomization, retinal correspondence status will be assessed by the Hering-Bielschowky after-image test, using a PEDIG-provided flash unit. Correspondence will be assessed when aligned and when tropic to record overall status as either:

IXT7ProtV1.0 19Apr2022 

| 620<br>621<br>622 | | Testing must be performed by a pediatric ophthalmologist, pediatric optometrist, or certified orthoptist as outlined in the <i>IXT7 Procedures Manual</i> . The examiner will be required to be masked to treatment group. Testing time is approximately 3-5 minutes. |
|---|---|---|
| 623<br>624<br>625<br>626<br>627<br>628<br>629<br>630<br>631<br>632<br>633<br>634<br>635<br>636 | 7. | Control of IXT: Assessment of IXT control will be performed using the Office Control Scale <sup>35</sup> at both distance (6 meters) and near (1/3 meter), fixating an accommodative target. Testing must be performed by a pediatric ophthalmologist, pediatric optometrist, or certified orthoptist as outlined in the IXT7 Procedures Manual. The examiner will be required to be masked to treatment group. Testing time is approximately 3-5 minutes. The scale below applies to both distance and near test distance separately. Intermittent Exotropia Control Scale 5 = Constant Exotropia 4 = Exotropia > 50% of the 30-second period before dissociation 3 = Exotropia < 50% of the 30-second period before dissociation 2 = No exotropia unless dissociated, recovers in >5 seconds 1 = No exotropia unless dissociated, recovers in 1-5 seconds 0 = No exotropia unless dissociated, recovers in <1 second (phoria) Not applicable = No exodeviation present |
| 638 | | Not applicable – No exodeviation present |
| 639 | | Directions: |
| 640 | | Step1: Assessment before any dissociation: Eye alignment is observed for a 30-second period |
| 641 | | with distance fixation. The time in seconds that a spontaneous IXT is observed is |
| 642 | | counted, and the appropriate control score (3, 4, or 5) is assigned for distance fixation. |
| 643 | | This is then repeated for near fixation for another 30-second period; if an exotropia is |
| 644 | | observed, then the time in seconds that an eye is observed to be exotropic is counted |
| 645 | | and the appropriate score of 3, 4, or 5 is assigned. If a score of $\geq$ 3 is present, then Step |
| 646 | | 2 (dissociation) is not required for that test distance. First distance and then near |
| 647 | | fixation are assessed before any dissociation (i.e., before step 2). |
| 648 | | Step 2: Assessment with standardized dissociation is performed only if spontaneous |
| 649 | | exotropia is NOT observed during step 1 (control was not a 3, 4, or 5). Instead, control |
| 650 | | will be a 0, 1, or 2; this is determined based on the worst score determined from 3 |
| 651 | | successive 10-second periods of dissociation: |
| 652 | | • An occluder is placed over the right eye for 10 seconds and then removed; the |
| 653 | | length of time it takes for the re-establishment of fusion is measured in seconds. |
| 654 | | • The left eye is then occluded for a 10-second period (second assessment under |
| 655 | | dissociation) and after uncovering the eye, the time for re-establishment of fusion |
| 656 | | is similarly measured in seconds. |
| 657 | | • A third assessment is performed, by covering the eye that required the longer time |
| 658 | | to re-fuse on the first two 10-second dissociations. After uncovering the eye, the |
| 659 | | length of time (in seconds) it takes for the reestablishment of fusion is measured |
| 660 | | in seconds. |

661662

should be recorded.

The worst level of control for the three 10-second periods of dissociation by occlusion

- Since the control score is the slowest time of the three assessments, if a score of 2 (>5 seconds recovery) is noted on the first or second dissociation, then subsequent dissociation(s) are not needed.
- If the child has a micro-esotropia by the cover-uncover test but an exodeviation by PACT, the control scale applies to the exodeviation.
  - 8. <u>Measurement of Divergence Amplitude:</u> Testing must be performed by a pediatric ophthalmologist, pediatric optometrist, or certified orthoptist. The examiner will be required to be masked to treatment group. Testing time is approximately 2-4 minutes.
    - Divergence amplitude to be measured at distance (6 meters)
    - Using the PEDIG-approved IXT7 prism bar, record the break, and recovery points according to the *IXT7 Testing Procedures Manual*.
    - If manifest exotropia is present at the time of testing, amplitude testing will be recorded as "unable."
  - 9. <u>Measurement of Convergence Amplitudes:</u> Testing must be performed by a pediatric ophthalmologist, pediatric optometrist, or certified orthoptist. The examiner will be required to be masked to treatment group. Testing time is approximately 2-4 minutes.
    - Convergence amplitude to be measured at distance (6 meters)
    - Using the PEDIG-approved IXT7 prism bar, record the blur, break, and recovery points according to the *IXT7 Testing Procedures Manual*.
    - If manifest exotropia is present at the time of testing, amplitude testing will be recorded as "unable."

The following information will be collected by interviewing the parent(s) or reviewing the medical record:

1) Date of birth, sex, race, ethnicity, spectacle correction, and prior treatment for IXT. Assessment of Adverse Events: All adverse events including ocular adverse events, and any events judged by the investigator to be related to patching treatment, occurring between the time of initiating study eye treatment and the 12-month outcome exam will be recorded.

Each questionnaire is described briefly below. The procedures for administration are described in the *IXT7 Testing Procedures Manual*.

# 1. Pediatric Eye Questionnaire (PedEyeQ)<sup>61</sup>

The Pediatric Eye Questionnaire (PedEyeQ), is a pediatric eye-related quality of life and functional vision instrument, validated for use in children with a variety of pediatric eye conditions. The PedEyeQ is patient- and parent-derived and consists of age-appropriate Child and Proxy components as well as a Parent component (to assess the effect on the parent themselves).

i. The Child PedEyeQ, designed for children 5 to 17 years, has the following 4 domains: Functional Vision, Bothered by Eyes and Vision. Social, and Frustration / Worry.

IXT7ProtV1.0 19Apr2022 

- ii. The Proxy PedEyeQ, designed for parents of children 0 to 17 years, has the following 5 domains: Functional Vision, Bothered by Eyes and Vision, Social, Frustration / Worry, and Eye care. Both the Child and Proxy PedEyeQ assess the eye-related quality of life and functional vision of the child.
- iii. The Parent PedEyeQ addresses the effect of the child's eye condition on the parent and has the following 4 domains: Impact on Parent and Family, Worry about Child's Eye Condition. Worry about Self-perception and Interactions, and Worry about Functional Vision.

Each of the Child, Proxy, and Parent domains is independently scored using established Rasch look-up tables and converted on a scale of 1 to 100 (each domain scored separately for each instrument). Completion time is approximately 10 minutes for the child, 10-15 minutes for the parent; child and parent questionnaires can be completed concurrently. The PedEyeQ questionnaires administered at enrollment will be the versions repeated throughout the study.

## 2. Intermittent Exotropia Symptom Survey<sup>62</sup>

The Intermittent Exotropia Symptom Survey is a patient- and parent-derived intermittent exotropia-related symptom instrument designed to identify the presence and severity of symptoms in children with IXT. This questionnaire consists of 22 items completed by children aged 5 years or older.

- All children will use the three-level response scale (not at all, sometimes, a lot), administered by clinical staff either verbally or using a matching card.
- If possible, children should be positioned such that they are unable to view their parents during testing and parents should be advised not to influence their child's responses.

Children 4 years and younger at enrollment will not complete the full questionnaire, but will answer the single question (#8) regarding diplopia. Time for completion of the full Symptom Survey is 5-7 minutes.

#### 3. Assessment of Diplopia by Parent

An estimate of the frequency of diplopia (if any) will be determined by asking the parent whether "your child has complained of double vision over the last week." If yes, the parent is asked how frequently the child has complained of double vision: "2 times or less per day," "or "more than 2 times per day." Any study personnel may ask the parent to rate diplopia. Testing time is approximately 1 minute.

IXT7ProtV1.0 19Apr2022 

## **Chapter 5: Unanticipated Problem and Adverse Event Reporting**

### **5.1 Unanticipated Problems**

744

745

750

751

752

753

754 755

756

757

758

759

760

761

762

763

764

765 766

- 746 Site investigators will promptly report to the Coordinating Center on an eCRF all unanticipated 747 problems meeting the criteria below. Sites must report Unanticipated Problems to the IRB within 748 seven (7) calendar days of recognition. For this protocol, an unanticipated problem is an incident, 749 experience, or outcome that meets all the following criteria:
  - Unexpected (in terms of nature, severity, or frequency) given (a) the research procedures that are described in the protocol related documents, such as the IRB-approved research protocol and informed consent document; and (b) the characteristics of the subject population being studied
  - Related or possibly related to participation in the research (possibly related means there is a reasonable possibility that the incident, experience, or outcome may have been caused by the procedures involved in the research)
  - Suggests that the research places participants or others at a greater risk of harm than was previously known or recognized (including physical, psychological, economic, or social

The Coordinating Center also will report to the IRB all unanticipated problems not directly involving a specific site such as unanticipated problems that occur at the Coordinating Center or at another participating entity such as a pharmacy or laboratory. These instances must be reported to the JCHR IRB within seven (7) calendar days of recognition. The Director of the Human Research Protection Program will report to the appropriate regulatory authorities if the IRB determines that the event indeed meets the criteria of an Unanticipated Problem that requires further reporting.

#### 767 768 **5.2 Adverse Events**

- 769 Although no adverse events are anticipated, any new reduction in VA of 3 or more lines (≥15 770 letters on ETDRS) or reduction in Randot Preschool Stereoacuity of 2 or more levels, will be
- 771 tabulated between treatment groups.
- 772 No surgical procedures are part of the protocol, and no treatments are being prescribed that are 773 not part of usual care. Investigators will abide by local IRB reporting requirements.

#### 774 **5.3 Safety Oversight**

- 775 A Data and Safety Monitoring Committee (DSMC) will review compiled safety data at periodic
- 776 intervals, with a frequency of no less than twice a year. The DSMC can request modifications to
- 777 the study protocol or suspension or outright stoppage of the study if deemed necessary based on
- 778 the totality of safety data available. Details regarding DSMC review will be documented in a 779 separate DSMC charter.
- 780 The objective of the DSMC review is to decide whether the study (or study treatment for an
- 781 individual or study cohort) should continue per protocol, proceed with caution, be further
- 782 investigated, be discontinued, or be modified and then proceed. Suspension of enrollment (for a
- 783 particular group, a particular study site, or for the entire study) is a potential outcome of a DSMC

784 safety review.

785

 IXT7PROTV1.0 19Apr2022

## 5.4 Stopping Criteria

- 787 The study may be discontinued by the Steering Committee (with approval of the Data and Safety
- 788 Monitoring Committee) prior to the preplanned completion of follow-up for all study
- participants. There are no pre-specified formal guidelines for stopping the study for futility or

790 efficacy.

791 792

794

795

796

799

786

## 5.5 Participant Discontinuation of Study Treatment

- Rules for discontinuing study treatment use are described below.
  - The investigator believes it is unsafe for the participant to continue to receive the treatment.
  - The participant or parent requests that the treatment be stopped.
- Even if the study treatment is discontinued, the participant will be encouraged to remain in the study through the 3-month visit.

IXT7ProtV1.0 19Apr2022 

| 800 | <b>Chapter 6: Miscellaneous Considerations</b> |
|---|---|
| 801 | 6.1 Contacts by the Jaeb Center for Health Research and Sites |
| 802<br>803 | The Jaeb Center serves as the PEDIG Coordinating Center. The Jaeb Center will be provided with the parent's contact information. The Jaeb Center may contact the parents of the |
| 804 | participants. Permission for such contacts will be included in the Informed Consent Form. The |
| 805 | principal purpose of the contacts will be to develop and maintain rapport with the participant and |
| 806 | family and to help coordinate scheduling of the outcome examinations. |
| 807 | (2 Participant Commonsation |
| 808<br>809 | 6.2 Participant Compensation Participant compensation will be specified in the informed consent form. |
| 810 | 6.3 Participant Withdrawal |
| | • |
| 811<br>812 | Participation in the study is voluntary, and a participant may withdraw at any time. For participants who withdraw, their data will be used up until the time of withdrawal. |
| 813 | 6.4 Confidentiality |
| 814<br>815<br>816<br>817 | For security and confidentiality purposes, participants will be assigned an identifier that will be used instead of their name. Protected health information gathered for this study will be shared with the coordinating center, the Jaeb Center for Health Research in Tampa, FL. De-identified participant information may also be provided to research sites involved in the study. |

IXT7ProtV1.0\_19Apr2022 

| 818 | <b>Chapter 7: Statistical Considerations</b> |
|---|---|
| 819<br>820<br>821 | 7.1 Statistical and Analytical Plans The approach to sample size and statistical analyses are summarized below. |
| 822<br>823 | <b>7.2 Primary Objective and Hypothesis</b> The study has one primary objective: |
| 824<br>825<br>826 | 1) To determine if participants with IXT undergoing full-time patching have more improvement in mean distance control between baseline and 3 months than participants being observed without treatment. |
| 827 | |
| 828<br>829 | The primary outcome is a comparison of the change in the mean distance control scores (average of 3 measurements) at 3 months between the full-time patching group and the observation group |
| 830<br>831<br>832 | The study is designed as a superiority study to evaluate two 2-sided primary null hypotheses that the changes in the mean control scores in the two groups at 3 months are the same versus the alternative hypothesis that they are different. |
| 833 | Hypothesis Test for Objective # 1 – FT vs OBS at 3 Months: |
| 834<br>835<br>836<br>837 | Hnull Halternative FT mean change in distance control over 3 months = OBS mean change in distance control over 3 months FT mean change in distance control over 3 months ≠ OBS mean change in distance control over 3 months |
| 838<br>839<br>840<br>841<br>842<br>843 | <b>7.3 Sample Size</b> Sample size estimation is based on data from our previous IXT2 randomized trial comparing observation versus part-time patching for intermittent exotropia, limited to 278 participants with similar baseline age (3 to <9 years) and baseline control score at distance (2 or higher). <sup>22</sup> Data are summarized in Table 1 below. |
| 844 | |

IXT7ProtV1.0\_19Apr2022 
Table 1 – Previous IXT2 Randomized Trial Data in 3- to <9-Year-Olds with IXT\*

| | Cohort | |
|---|---|---|
| | IXT2<br>Glasses Alone | IXT2 Part-time Patching |
| Distance Control Scores** | (Observation) | (3 hours/Day) |
| Baseline | | |
| n | 147 | 131 |
| Mean (SD) | 2.88 (1.01) | 2.93 (1.00) |
| 3-Month Score | | |
| n | 131 | 116 |
| Mean Score (SD) | 2.59 (1.35) | 2.15 (1.23) |
| 95% CI for Mean Score | 2.35 to 2.82 | 1.92 to 2.37 |
| 95% CI for SD Score | 1.21 to 1.54 | 1.09 to 1.41 |
| 3-Month Change from Baseline | | |
| n | 131 | 116 |
| Mean Change (SD) | 0.30 (1.23) | 0.78 (1.38) |
| 95% CI for Mean Change | 0.09 to 0.51 | 0.53 to 1.04 |
| 95% CI for SD Change | 1.09 to 1.40 | 1.22 to 1.59 |

<sup>\*</sup>Participants aged 3 to <9 years old with baseline distance control score of 2 or higher (worse).

In IXT2, after 3 months of observation versus treatment with 3 hours per day patching, the observation group had a mean change based upon a single measure of distance control of 0.30 points (95% CI, 0.09 to 0.51 points) with a standard deviation of 1.23 points (95% CI, 1.09 to 1.40 points); and the 3 hours per day patching group had a mean change based upon a single measure of distance control of 0.78 points (95% CI, 0.53 to 1.04 points) with a standard deviation of 1.38 points (95% CI, 1.22 to 1.59 points); group difference patching – observation = 0.49 (95% CI 0.16 to 0.81). The correlation between distance control score at baseline and change from baseline after 3 months was R=0.39 (95% CI, 0.27 to 0.48).

We are aware of no previous data on distance control score among children with IXT treated with full-time patching. In our IXT5 study, after 6 months of treatment with overminus spectacles, the mean change in distance control was 1.40 points (95% CI, 1.18 to 1.63 points) with a standard deviation of 1.48 points (95% CI, 1.34 to 1.66 points). There was no 3-month outcome in the IXT5 study; however, in the IXT3 pilot study, those treated with overminus spectacles improved on average 1.2 points (95% CI, 0.5 to 1.9 points) with a standard deviation of 1.8 points (95% CI, 1.4 to 2.5 points) after 8 weeks. Therefore, we estimate that a mean change of 1.45 points after 3 months of full-time patching in the current study is reasonable for an active treatment.

#### **Sample Size Estimation:**

- The study will be powered for the primary objective.
- Assuming a mean change in distance control score after 3 months of 0.30 points in the observation group and 1.45 points in the full-time patching group; we estimate that the true difference is 1.15 points between full-time patching and observation at 3 months.

<sup>\*\*</sup> A single measure of control was obtained at each visit in the IXT2 study.

#### **Hypothesis Test for Objective – FT vs OBS at 3 Months:**

Assuming a pooled standard deviation of 1.5 points for change in distance control score after 3 874 875 months, and a correlation of 0.30 between distance control score at baseline and change from

876 baseline after 3 months, a total sample size of 68 participants (34 per group) completing the 3-

month outcome has 90% power with a type I error rate of 5% to evaluate whether there is a 877

treatment group difference between FT patching and OBS if the true difference is 1.15 points. 878

879 Table 2. Accounting for 5% loss to follow-up after 3 months, a total of 72 participants (36 per

880 treatment group) will need to be enrolled. The overall number of participants with an interocular

881 difference in distance VA of 2 logMAR lines (10 letters on E-ETDRS for patients ≥7 years old) will be

882 limited to 14.

## Table 2: Total Sample Size for Difference in Mean Distance Control Score

| <b>Standard Deviation</b> | Treatment Group I | Difference for Outcome | of Mean Change in |
|---|---|---|---|
| of Change in Distance | Distance Control (points) | | |
| Control (points) | 0.85 | 1.00 | 1.15 |
| 1.4 | 106 | 78 | 60 |
| 1.5 | 122 | 90 | 68 |
| 1.6 | 138 | 100 | 78 |

Cells indicate N for the overall study (two treatment groups combined with a ratio of 1:1), using a 2-sided test with alpha 0.05, from an analysis of covariance model evaluating a difference between treatment groups for mean change from baseline in distance control, controlling for baseline distance control.

887

888

889

890

891 892

893

896

897

898

899

900

901

902

903

904

905

884

885

886

873

883

If the true effect with FT patching is as small as 0.99, the study would still have 80% power to reject the null in favor of a difference (and 1.05 with 85%).

## 7.4 Interim Monitoring

Given the short duration of the primary outcome at 3 months, there will be no formal interim analysis for stopping the study early for efficacy or futility.

#### 7.5 Analysis Datasets

894 The primary efficacy analysis will follow an intent-to-treat (ITT) principle. Therefore, the 895 primary analysis dataset will include all randomized participants with imputation for those missing the 3-month outcome and will analyze them according to the group they were originally assigned. Sensitivity analyses of the primary outcome will follow a modified ITT principle and use observed data with no imputation for missing outcomes.

#### 7.6 Analysis of the Primary Efficacy Endpoints

The mean of three individual distance control scores will be tabulated by treatment group at 3 months. The change from baseline in mean control score (mean of three assessments) will be compared between the FT patching group and the OBS group at 3 months using an analysis of covariance (ANCOVA) model that adjusts for the mean distance control score at baseline and distance angle by PACT at baseline. An estimate of difference between the groups will be reported along with a 95% confidence interval and p-value.

 IXT7ProtV1.0 19Apr2022

- When the protocol-specified three measures of control are not performed at the outcome exam,
- the mean of two tests will be used for analysis if only 2 distance control tests are completed; the
- single distance control score will be used for analysis if only 1 testing is completed.
- Participants who miss the 3-month visit or who do not complete any control testing at the 3-
- 910 month visit will have an average distance control score imputed using multiple imputation.
- The multiple imputation will be performed using Monte Carlo Markov Chain (MCMC) modeling
- that includes the mean distance controls at the outcome visit and the following baseline factors:
- 913 mean distance control, and distance PACT.

## 914 **7.6.1 Sensitivity Analyses**

- The following analyses will be performed as sensitivity analyses to the primary analysis:
- 916 Sensitivity Analysis #1 (Complete Case Analysis Including Visits within Analysis Window):
- All participants who complete 1 or more distance control tests at the 3-month visit within the analysis window (± 1 month) will have their observed 3-month data analyzed
- Participants who miss the 3-month visit entirely or who do not complete any control testing at the 3-month visit within the analysis window will be excluded from the analysis
- 921 Sensitivity Analysis #2 (Complete Case Analysis Including Visits within Protocol Window):
- Repeat the above sensitivity analysis using observed data from participants who completed the 3-month visit within the protocol window (± 2 weeks).
- 925 Sensitivity Analysis #3 (ITT minus participants with IOD 2 logMAR lines at enrollment):
- The overall number of participants with an interocular difference in distance VA of 2
   logMAR lines (10 letters on E-ETDRS for patients ≥7 years old) will be limited to 14.
- The ITT analyses as described in 7.5 will be repeated excluding these participants.

#### 930 7.7 Analysis of the Secondary Endpoints

- All secondary analyses described below will use observed data only. Treatment group
- comparisons specified in the sections below will be controlled using false discovery rate (FDR)
- at the 5% probability level to account for the multiple outcomes. For all secondary analyses, an
- estimate of difference between the groups will be reported at each timepoint along with an FDR-
- adjusted confidence interval and p-value unless otherwise specified. Further details about the
- 936 secondary analyses below will be part of a separate statistical analysis plan (SAP).

#### 937 **7.7.1 Near Control**

924

929

- At 3 months, near control will be evaluated similarly to the distance control primary analysis
- 939 (section 7.6) using ANCOVA models that adjust for the mean near control score at baseline and
- 940 the near angle by PACT at baseline.
- Additionally, the proportion of participants with 2 or more points improvement in control from
- baseline will be compared between the treatment groups at 3 months using a two-sided Barnard's
- 943 test with calculation of a two-sided FDR-adjusted confidence interval on the difference in
- proportions. This will be done separately for control at distance and near.

IXT7ProtV1.0 19Apr2022 

| 945 <b>7.7.2 Angle of Deviation</b> | 945 | 7.7.2 | Angle | of Dev | viatior |
|-------------------------------------|-----|-------|-------|--------|---------|
|-------------------------------------|-----|-------|-------|--------|---------|

- At 3 months, a two-sided comparison of magnitude of the angle of deviation by PACT will be
- 947 performed between treatment groups using an ANCOVA model, which adjusts for baseline
- 948 PACT. The treatment group difference and an FDR-adjusted confidence interval will be
- calculated. The analysis will be completed separately at distance and at near.
- Additionally, the proportion of participants with improvement of distance and near angle greater
- than the test/retest variability<sup>63</sup> will be compared between the treatment groups at 3 months using
- a two-sided Barnard's test with calculation of a two-sided FDR-adjusted confidence interval on
- 953 the difference in proportions.

## 954 7.7.3 Level of Suppression

- The proportion with each level of suppression (negligible, mild, moderate, or dense) will be
- compared between treatment groups at 3 months using an exact Wilcoxon rank sum test.

## 957 7.7.4 Proportion with Anomalous Retinal Correspondence

- 958 For those able to perform the test, the proportions of normal versus anomalous retinal
- orrespondence will be compared between treatment groups at 3 months using a two-sided
- 960 Barnard's test for the difference in proportions.

## 961 7.7.5 Convergence and Divergence Fusional Amplitudes

- The distribution of fusional convergence amplitude (blur point, break point, and recovery) and
- 963 fusional divergence amplitude (break point and recovery point) will be described and compared
- between treatment groups at 3 months using an exact Wilcoxon rank sum test. When no blur is
- reported for fusion convergence, the break point will be used for analysis.

#### 966 7.7.6 IXT Symptom Survey Score

- The IXT Symptom Survey will be completed by children at the enrollment and 3-month exams.
- The distribution for each individual item ('Never', 'Sometimes', 'All the Time) will be tabulated
- 969 for each treatment group within subgroups defined by age 5 to 9 years (all items) and age <5
- years for the single diplopia question.

#### **7.7.7 PedEveQ Score**

- The PedEyeQ consists of 3 components: child, proxy, and parent. After applying existing Rasch
- scoring, 61 the average score for each of the domains within the three components will be
- ompared between treatment groups at 3 months using an ANCOVA model, which adjusts for
- baseline PedEveO score. The treatment group difference and an FDR-adjusted confidence
- 976 interval will be calculated.

## 977 7.7.8 Binocular Diplopia by Parental Report

- The proportion of binocular diplopia at 3 months with a frequency of "more than 2 times per
- day" over the last week at distance or near, by parental report will be compared treatment groups
- at 3 months using a two-sided Barnard's test.

981

IXT7ProtV1.0 19Apr2022 

| 982 | 7.8 Exploratory Analyses |
|---|---|
| 983<br>984 | Exploratory analyses described below will use observed data only. Point estimates and 95% CIs will be reported for each outcome with no adjustment for multiplicity. |
| 985<br>986<br>987<br>988 | <b>7.8.1 Actual Patch Wear Time</b> The distribution of actual patch wear time will be tabulated overall and by treatment groups. The potential correlation between actual patch wear time in the FT patching group and the change from baseline in the following outcomes will be evaluated at 3 months (when collected): |
| 989<br>990<br>991<br>992<br>993<br>994<br>995<br>996<br>997 | <ol> <li>Distance control score</li> <li>Near control score</li> <li>Distance angle of deviation</li> <li>Near angle of deviation</li> <li>Level of suppression</li> <li>Convergence fusional amplitudes</li> <li>Divergence fusional amplitudes</li> <li>Symptom survey score</li> <li>Diplopia assessment by Parent</li> <li>PedEyeQ score (each domain)</li> </ol> |
| 999<br>1000 | A Spearman correlation coefficient and 95% confidence interval will be calculated for each outcome. |
| 1001<br>1002<br>1003 | <b>7.8.2 Outcome of Retinal Correspondence Testing</b> The relationship of retinal correspondence response with respect to the following outcomes within each treatment group will be evaluated at 3 months: |
| 1004<br>1005<br>1006<br>1007<br>1008<br>1009<br>1010<br>1011<br>1012 | <ol> <li>Distance control score</li> <li>Near control score</li> <li>Distance angle of deviation</li> <li>Near angle of deviation</li> <li>Level of suppression</li> <li>Convergence fusional amplitudes</li> <li>Divergence fusional amplitudes</li> <li>Symptom survey score</li> <li>Diplopia assessment by Parent</li> <li>PedEyeQ score</li> </ol> |
| 1014<br>1015<br>1016<br>1017 | For continuous outcome variables, the difference in means between participants with normal versus anomalous retinal correspondence will be calculated along with a 95% confidence interval. For categorical outcome variables, the difference in proportions between participants with normal versus anomalous retinal correspondence will be calculated along with a 95% confidence interval. |

IXT7ProtV1.0\_19Apr2022 

7.8.3 Subgroup Analysis of Distance Control

1019

| 1020<br>1021<br>1022<br>1023 | The treatment group comparison of distance control will be assessed at 3 months in subgroups based on gender and race/ethnicity in accordance with NIH guidelines; however, no effect modification is expected for these factors. |
|---|---|
| 1024 | 7.9 Safety Analyses |
| 1025 | |
| 1026<br>1027<br>1028 | <b>7.9.1 Deterioration</b> The number and proportion of participants with deterioration, as defined below, will be tabulated for each treatment group at 3 months as a safety outcome. |
| 1029<br>1030 | Deterioration is defined as meeting one of the following criteria at the 3 months follow-up visit: |
| 1031<br>1032<br>1033<br>1034<br>1035<br>1036 | <ol> <li>Constant exotropia at least 10Δ at distance AND near by SPCT: <ul> <li>Constant is defined as an exotropia present throughout the examination and confirmed by cover/uncover testing performed at least 3 different times over the course of the exam (including during assessment of IXT control).</li> </ul> </li> <li>Decrease in near stereoacuity of at least 2 levels from baseline, or to nil, measured using the Randot Preschool Stereotest.</li> </ol> |
| 1037<br>1038<br>1039<br>1040 | <b>7.9.2 Reduction of Distance Visual Acuity</b> Any cases of 1) interocular difference ≥0.3 logMAR and 2) reduced visual acuity in best refractive correction (≥0.3 logMAR) in either eye will be tabulated by treatment group at 3 months. |
| 1041 | 7.9.3 Diplopia |
| 1042<br>1043<br>1044<br>1045<br>1046 | After 3 months, any new cases of diplopia 'Sometimes' or 'All the Time', based on response to item 8 from the IXT symptom survey (asked as a single question for children ages 3 and 4 years of age) will be tabulated for each treatment group. In addition, diplopia occurring 'Never', 'Sometimes', or 'All the Time' will also be tabulated for each treatment group. |
| 1047 | 7.10 Patching Adherence |
| 1048<br>1049 | Patching adherence (as reported by the parent) will be tabulated at the 3-month visit for the FT patching treatment group, as will reasons for any major deviations. |
| 1050<br>1051<br>1052<br>1053<br>1054<br>1055<br>1056 | <ul> <li>7.11 Additional Tabulations and Analyses</li> <li>The following tabulations and analyses will be performed: <ul> <li>A flow chart accounting for all participants according to treatment group</li> <li>Visit completion rates according to treatment group</li> <li>Baseline demographics and clinical characteristics overall and by treatment group at randomization</li> <li>Protocol deviations according to treatment group</li> </ul> </li> </ul> |

IXT7ProtV1.0\_19Apr2022 

#### **Chapter 8: Data Collection and Monitoring** 1057

#### 8.1 Case Report Forms and Other Data Collection

- 1059 The main study data are collected on electronic case report forms (CRFs). When data are directly
- 1060 collected in electronic case report forms, this will be considered the source data. For any data
- points for which the eCRF is not considered source (e.g., lab results that are transcribed from a 1061
- 1062 printed report into the eCRF), the original source documentation must be maintained in the
- participant's study chart or medical record. This source must be readily verifiable against the 1063
- 1064 values entered into eCRF. Even where all study data are directly entered into the eCRFs at office
- 1065 visits, evidence of interaction with a live participant must be recorded (e.g., office note, visit
- record, etc.). 1066

1058

1072 1073

1074

1075

1079 1080

- 1067 Electronic device data files are obtained from the study software and individual hardware
- 1068 components. These electronic device files are considered the primary source documentation.
- 1069 Each participating site will maintain appropriate medical and research records for this trial, in
- 1070 compliance with ICH E6 and regulatory and institutional requirements for the protection of
- 1071 confidentiality of participants.

## **8.2 Study Records Retention**

Study documents should be retained for a minimum of 3 years after completion of the final grant reporting. These documents should be retained for a longer period, however, if required by local

1076 regulations. No records will be destroyed without the written consent of the sponsor, if

1077 applicable. It is the responsibility of the sponsor to inform the investigator when these documents 1078

no longer need to be retained.

## **8.3 Quality Assurance and Monitoring**

- 1081 Designated personnel from the Coordinating Center will be responsible for maintaining quality
- 1082 assurance (QA) and quality control (QC) systems to ensure that the clinical portion of the trial is
- 1083 conducted and data are generated, documented and reported in compliance with the protocol
- 1084 adhering to Good Clinical Practice (GCP) and the applicable regulatory requirements, as well as
- to ensure that the rights and wellbeing of trial participants are protected and that the reported trial 1085
- data are accurate, complete, and verifiable. Adverse events will be prioritized for monitoring. 1086
- 1087 A risk-based monitoring (RBM) plan will be developed and revised as needed during the course
- 1088 of the study, consistent with the FDA "Guidance for Industry Oversight of Clinical
- 1089 Investigations — A Risk-Based Approach to Monitoring" (August 2013). This plan describes in
- 1090 detail who will conduct the monitoring, at what frequency monitoring will be done, at what level
- 1091 of detail monitoring will be performed, and the distribution of monitoring reports.
- 1092 The data of most importance for monitoring at the site are participant eligibility and adverse
- 1093 events. Therefore, the RBM plan will focus on these areas. As much as possible, remote
- 1094 monitoring will be performed in real-time with on-site monitoring performed to evaluate the
- 1095 verity and completeness of the key site data.

1096

 IXT7ProtV1.0 19Apr2022

## 1097 Elements of the RBM may include:

- Qualification assessment, training, and certification for sites and site personnel
- Oversight of Institutional Review Board (IRB) coverage and informed consent procedures
  - Central (remote) data monitoring: validation of data entry, data edits/audit trail, protocol review of entered data and edits, statistical monitoring, study closeout
  - On-site monitoring (site visits): source data verification, site visit report
- Agent/Device accountability
  - Communications with site staff
  - Patient retention and visit completion
- Quality control reports
- Management of noncompliance
- Documenting monitoring activities
- Adverse event reporting and monitoring
- 1111 Coordinating Center representatives or their designees may visit the study facilities at any time in
- order to maintain current and personal knowledge of the study through review of the records,
- 1113 comparison with source documents, observation and discussion of the conduct and progress of
- the study. The investigational site will provide direct access to all trial related sites, source
- data/documents, and reports for the purpose of monitoring and auditing by the sponsor, and
- inspection by local and regulatory authorities.

## 1117

1098

1101 1102

1103

1105

1106

- 1118 **8.4 Protocol Deviations**
- 1119 A protocol deviation is any noncompliance with the clinical trial protocol, GCP, or procedure
- requirements. The noncompliance may be either on the part of the participant, the investigator, or
- the study site staff. As a result of deviations, corrective actions are to be developed by the site
- and implemented promptly.
- The site PI/study staff is responsible for knowing and adhering to their IRB requirements.
- Further details about the handling of protocol deviations will be included in the monitoring plan.

IXT7ProtV1.0 19Apr2022 

# Chapter 9: Ethics/Protection of Human Participants

#### 1126 9.1 Ethical Standard

- The investigator will ensure that this study is conducted in full conformity with Regulations for
- the Protection of Human Participants of Research codified in 45 CFR Part 46, 21 CFR Part 50,
- 1129 21 CFR Part 56, and/or the ICH E6.

## 1130 1131

1125

#### 9.2 Institutional Review Boards

- The protocol, informed consent form(s), recruitment materials, and all participant materials will
- be submitted to the IRB for review and approval. Approval of both the protocol and the consent
- form must be obtained before any participant is enrolled. Any amendment to the protocol will
- require review and approval by the IRB before the changes are implemented to the study. All
- changes to the consent form will be IRB approved; a determination will be made regarding
- whether previously consented participants need to be re-consented.

## 1138 1139

1140

1157

#### 9.3 Informed Consent Process

#### 9.3.1 Consent Procedures and Documentation

- Informed consent is a process that is initiated prior to the individual's agreeing to participate in
- the study and continues throughout the individual's study participation. Extensive discussion of
- risks and possible benefits of participation will be provided to the participants and their families.
- 1144 Consent forms will be IRB-approved and the participant will be asked to read and review the
- document. The investigator will explain the research study to the participant and answer any
- 1146 questions that may arise. All participants will receive a verbal explanation in terms suited to their
- 1147 comprehension of the purposes, procedures, and potential risks of the study and of their rights as
- research participants. Participants will have the opportunity to carefully review the written
- 1149 consent form and ask questions prior to signing.
- The participants should have the opportunity to discuss the study with their surrogates or think
- about it prior to agreeing to participate. The participant will sign the informed consent document
- prior to any procedures being done specifically for the study. The participants may withdraw
- 1153 consent at any time throughout the course of the trial. A copy of the informed consent document
- will be given to the participants for their records. The rights and welfare of the participants will
- be protected by emphasizing to them that the quality of their medical care will not be adversely
- affected if they decline to participate in this study.

#### 9.3.2 Participant and Data Confidentiality

- Participant confidentiality is strictly held in trust by the participating investigators, their staff,
- and the sponsor(s) and their agents. This confidentiality is extended to cover testing of biological
- samples and genetic tests in addition to the clinical information relating to participants.
- Therefore, the study protocol, documentation, data, and all other information generated will be
- held in strict confidence. No information concerning the study or the data will be released to any
- unauthorized third party without prior written approval of the sponsor.
- The study monitor, other authorized representatives of the sponsor, representatives of the IRB,
- regulatory agencies or company supplying study product may inspect all documents and records
- required to be maintained by the investigator, including but not limited to, medical records

IXT7ProtV1.0 19Apr2022 

- 1167 (office, clinic, or hospital) and pharmacy records for the participants in this study. The clinical
- study site will permit access to such records.
- The study participant's contact information will be securely stored at each clinical site for
- internal use during the study. At the end of the study, all records will continue to be kept in a
- secure location for as long a period as dictated by the reviewing IRB, institutional policies, or
- sponsor requirements.
- 1173 Study participant research data, which is for purposes of statistical analysis and scientific
- reporting, will be transmitted to and stored at the Jaeb Center for Health Research. This will not
- include the participant's contact or identifying information. Rather, individual participants and
- their research data will be identified by a unique study identification number. The study data
- entry and study management systems used by clinical sites and by Jaeb Center for Health
- Research staff will be secured and password protected.
- 1179 At the end of the study, all study databases will be de-identified and archived at the Jaeb Center
- 1180 for Health Research.
- To further protect the privacy of study participants, a Certificate of Confidentiality will be
- obtained from the NIH. This certificate protects identifiable research information from forced
- disclosure. It allows the investigator and others who have access to research records to refuse to
- disclose identifying information on research participation in any civil, criminal, administrative,
- legislative, or other proceeding, whether at the federal, state, or local level. By protecting
- researchers and institutions from being compelled to disclose information that would identify
- research participants, Certificates of Confidentiality help achieve the research objectives and
- promote participation in studies by helping assure confidentiality and privacy to participants.
- 1189 **9.3.3 Future Use of Data**
- Data collected for this study will be analyzed and stored at the Jaeb Center for Health Research.
- After the study is completed, the de-identified, archived data will be made available to the
- 1192 public.

IXT7ProtV1.0 19Apr2022 

# **Chapter 10: References**

- 1193
- 1. Govindan M, Mohney BG, Diehl NN, Burke JP. Incidence and types of childhood exotropia: A population-based study. *Ophthalmology*. 2005;112(1):104-108.
- Friedman DS, Repka MX, Katz J, et al. Prevalence of amblyopia and strabismus in white and African American children aged 6 through 71 months. The Baltimore Pediatric Eye Disease Study. *Ophthalmology*. 2009;116(11):2128-2134.
- Nusz KJ, Mohney BG, Diehl NN. Female predominance in intermittent exotropia. *Am J Ophthalmol.* 2005;140(3):546-547.
- 1201 4. Chia A, Dirani M, Chan YH, et al. Prevalence of amblyopia and strabismus in young singaporean chinese children. *Invest Ophthalmol Vis Sci.* 2010;51(7):3411-3417.
- 1203 5. Chia A, Roy L, Seenyen L. Comitant horizontal strabismus: an Asian perspective. *Br J Ophthalmol.* 2007;91(10):1337-1340.
- 1205 6. McKean-Cowdin R, Cotter SA, Tarczy-Hornoch K, et al. Prevalence of amblyopia or strabismus in Asian and non-Hispanic white preschool children: Multi-ethnic Pediatric Eye Disease Study. *Ophthalmology*. 2013;120(10):2117-2124.
- 7. Costenbader F. The physiology and mangement of divergent strabismus. In: Allen JH, ed. Strabismic ophthalmic symposium. St. Louis: Mosby Year Book; 1950:353.
- Burian HM, Smith DR. Comparative measurement of exodeviations at twenty and one hundred feet. *Trans Am Ophthalmol Soc.* 1971;69:188-199.
- 1212 9. Cooper J. Intermittent exotropia of the divergence excess type. *J Am Optom Assoc*. 1213 1977;48(10):1261-1273.
- 1214 10. Campos EC, Cipolli C. Binocularity and photophobia in intermittent exotropia. *Percept* 1215 *Mot Skills*. 1992;74(3 pt 2):1168-1170.
- 1216 11. Wang FM, Chryssanthou G. Monocular eye closure in intermittent exotropia. *Arch Ophthalmol.* 1988;106(7):941-942.
- 1218 12. Wiggins RE, von Noorden GK. Monocular eye closure in sunlight. *J Pediatr Ophthalmol Strabismus*. 1990;27(1):16-20.
- 1220 13. Hatt SR, Leske DA, Mohney BG, Brodsky MC, Holmes JM. Classification and
   1221 misclassification of sensory monofixation in intermittent exotropia. *Am J Ophthalmol*.

1222 2010;150(1):16-22.

- 1223 14. Hatt S, Gnanaraj L. Interventions for intermittent exotropia. *Cochrane Database Syst* 1224 *Rev.* 2013(5):Art. No.: SAHA02.
- 1225 15. Pratt-Johnson JA, Barlow JM, Tillson G. Early surgery in intermittent exotropia. *Am J Ophthalmol*. 1977;84(5):689-694.
- 1227 16. Cooper J, Medow N. Intermittent exotropia, basic and divergence excess type. *Binocular Vision & Strabismus Quarterly*. 1993;8(3):187-216.
- 1230 Serrano-Pedraza I, Manjunath V, Osunkunle O, Clarke MP, Read JC. Visual suppression in intermittent exotropia during binocular alignment. *Invest Ophthalmol Vis Sci.* 2011;52(5):2352-2364.
- 1232 18. Cooper J, Record CD. Suppression and retinal correspondence in intermittent exotropia.

  1233 Br J Ophthalmol. 1986;70(9):673-676.
- 1234 19. Cooper J, Feldman J. Panoramic viewing, visual acuity of the deviating eye, and anomalous retinal correspondence in the intermittent exotrope of the divergence excess type. *Am J Optom Physiol Opt.* 1979;56(7):422-429.

IXT7ProtV1.0 19Apr2022 

- 1237 20. Romano PE, Wilson MF. Survey of current management of intermittent exotropia in the
   1238 USA and Canada. In: Campos EC, ed. *Strabismus and Ocular Motility Disorders*.
   1239 London: The Macmillan Press; 1990:391-396.
- Barnett-Itzhaki G, Friehmann A, Barnett-Itzhaki Z, Ela-Dalman N. Diagnosis and
   Management Practice Patterns among Pediatric Ophthalmology Personnel in Israel. J
   Binocul Vis Ocul Motil. 2019;69(1):34-41.
- Pediatric Eye Disease Investigator Group. A randomized trial comparing part-time patching with observation for children 3 to 10 years of age with intermittent exotropia. *Ophthalmology.* 2014;121(12):2299-2310.
- Pediatric Eye Disease Investigator Group. A randomized trial comparing part-time patching with observation for intermittent exotropia in children 12 to 35 months of age. *Ophthalmology*. 2015;122(8):1718-1725.
- Mohney BG, Cotter SA, Chandler DL, et al. Three-year observation of children 3 to 10 years of age with untreated intermittent exotropia. *Ophthalmology*. 2019;126(9):1249-1251 1260.
- Holmes JM, Hercinovic A, Melia BM, et al. Health-related quality of life in children with untreated intermittent exotropia and their parents. *J AAPOS*. 2021;25(2):80.e81-80.e84.
- Cotter SA, Mohney BG, Chandler DL, et al. Three-year observation of children 12 to 35 months old with untreated intermittent exotropia. *Ophthalmic Physiol Opt.* 2020;40(2):202-215.
- 1257 27. Clarke M, Hogan V, Buck D, et al. An external pilot study to test the feasibility of a 1258 randomised controlled trial comparing eye muscle surgery against active monitoring for 1259 childhood intermittent exotropia [X(T)]. *Health Technol Assess*. 2015;19(39):1-144.
- Pediatric Eye Disease Investigator Group. A randomized trial comparing bilateral lateral rectus recession versus unilateral recess and resect for basic-type intermittent exotropia.

  Ophthalmology. 2019;126(2):305-317.
- 1263 29. Kushner BJ. Selective surgery for intermittent exotropia based on distance/near differences. *Arch Ophthalmol*. 1998;116(3):324-328.
- Repka MX, Chandler DL, Holmes JM, et al. The Relationship of Age and Other Baseline
   Factors to Outcome of Initial Surgery for Intermittent Exotropia. *Am J Ophthalmol*.
   2020;212:153-161.
- 1268 31. Chen AM, Erzurum SA, Chandler DL, et al. Overminus lens therapy for children 3 to 10 years of age with intermittent exotropia: A randomized clinical trial. *JAMA Ophthalmol*. 2021;139(4):464-476.
- 1271 32. Flynn JT, McKenney S, Rosenhouse M. Management of intermittent exotropia. In:
- Moore S, Mein J, Stockbridge L, eds. *Orthoptics: Past, Present, Future*. Chicago: Year Book Medical Publishers; 1976:551-557.
- 1274 33. Iacobucci I, Henderson JV. Occlusion in the preoperative treatment of exotropia. *Am Orthopt J.* 1965;15:42-47.
- 1276 34. Akbari MR, Mehrpour M, Mirmohammadsadeghi A. The influence of alternate part-time patching on control of intermittent exotropia: a randomized clinical trial. *Graefes Arch Clin Exp Ophthalmol.* 2021;259(6):1625-1633.
- 1279 35. Mohney BG, Holmes JM. An office-based scale for assessing control in intermittent exotropia. *Strabismus*. 2006;14(3):147-150.
- 1281 36. Coffey B, Wick B, Cotter S, Scharre J, Horner D. Treatment options in intermittent exotropia: a critical appraisal. *Optom Vis Sci.* 1992;69(5):386-404.

IXT7ProtV1.0 19Apr2022 

- Heydarian S, Hashemi H, Jafarzadehpour E, et al. Non-surgical management options of intermittent exotropia: A literature review. *J Curr Ophthalmol*. 2020;32(3):217-225.
- 1285 38. AlKahmous LS, Al-Saleh AA. Does occlusion therapy improve control in intermittent exotropia? *Saudi Journal of Ophthalmology*. 2016;30(4):240-243.
- 1287 39. Kushner BJ. Conservative management of intermittent exotropia to defer or avoid surgery. *J AAPOS*. 2019;23(5):256.e251-256.e256.
- 1289 40. Jampolsky A. Physiology of intermittent exotropia. *Am Orthopt J.* 1963;13:5-13.
- 1290 41. Pratt-Johnson J, Wee HS. Suppression associated with exotropia. *Can J Ophthalmol*. 1291 1969;4(2):136-144.
- 1292 42. Cooper J, Feldman J, Pasner K. Intermittent exotropia: stimulus characteristics affect tests for retinal correspondence and suppression. *Binocul Vis Strabismus Q*. 2000;15(2):131-140.
- 1295 43. Yildirim C, Altinsoy HI. Distance alternate-letter suppression test for objective 1296 assessment of sensorial status in intermittent exotropia. *Eur J Ophthalmol*. 2000;10(1):4-1297 10.
- Wakayama A, Nakada K, Abe K, Matsumoto C, Shimomura Y. Effect of suppression during tropia and phoria on phoria maintenance in intermittent exotropia. *Graefes Arch Clin Exp Ophthalmol*. 2013;251(10):2463-2469.
- Hatt SR, Leske DA, Mohney BG, Brodsky MC, Holmes JM. Fusional convergence in childhood intermittent exotropia. *Am J Ophthalmol.* 2011;152:314-319.
- 1303 46. Liebermann L, Hatt SR, Leske DA, et al. Assessing divergence in children with intermittent exotropia. *Strabismus*. 2012;20(1):11-16.
- 1305 47. Chutter CP. Occlusion treatment of intermittent divergent strabismus. *Am Orthopt J.* 1306 1977;27:80-84.
- 1307 48. Vishnoi SK, Singh V, Mehra MK. Role of occlusion in treatment of intermittent exotropia. *Indian J Ophthalmol*. 1987;35(4):207-210.
- 1309 49. Spoor DK, Hiles DA. Occlusion therapy for exodeviations occurring in infants and young children. *Ophthalmology*. 1979;86(12):2152-2157.
- Bang SP, Lee DC, Lee SY. Surgical outcome of intermittent exotropia with improvement in control grade subsequent to part-time preoperative occlusion therapy. *J Pediatr Ophthalmol Strabismus*. 2018;55(1):59-64.
- Wang J, Xu H, De La Cruz B, et al. Improved monitoring of adherence with patching treatment using a microsensor and Eye Patch Assistant. *J AAPOS*. 2020;24(2):94.e91-94.e97.
- Fielder AR, Irwin M, Auld R, Cocker KD, Jones HS, Moseley MJ. Compliance in amblyopia therapy: objective monitoring of occlusion. *Br J Ophthalmol*. 1995;79(6):585-589.
- Stewart CE, Stephens DA, Fielder AR, Moseley MJ, ROTAS Cooperative. Objectively monitored patching regimens for treatment of amblyopia: randomised trial. *Br Med J*. 2007;335(7622):707-713.
- Loudon SE, Passchier J, Chaker L, et al. Psychological causes of non-compliance with electronically monitored occlusion therapy for amblyopia. *Br J Ophthalmol*. 2009;93(11):1499-1503.
- Holmes JM, Hercinovic A, Melia BM, et al. Health-related quality of life in children with untreated intermittent exotropia and their parents. *J AAPOS*. 2021.

IXT7ProtV1.0 19Apr2022 

- 1328 56. Drover JR, Felius J, Cheng CS, Morale SE, Wyatt L, Birch EE. Normative pediatric visual acuity using single surrounded HOTV optotypes on the Electronic Visual Acuity Tester following the Amblyopia Treatment Study protocol. *J AAPOS*. 2008;12(2):145-1331 149.
- Pan Y, Tarczy-Hornoch K, Cotter SA, et al. Visual acuity norms in pre-school children: the Multi-Ethnic Pediatric Eye Disease Study. *Optom Vis Sci.* 2009;86(6):607-612.
- Morale SE, Cheng-Patel CS, Jost RM, Donohoe N, Leske DA, Birch EE. Normative
   pediatric visual acuity using electronic Early Treatment for Diabetic Retinopathy protocol
   *J AAPOS*. 2021;25(3):172-175.
- Hatt SR, Leske DA, Holmes JM, et al. Testing depth of suppression in childhood intermittent exotropia. *J aapos*. 2021.
- 1339 60. Bielschowsky A. Divergence excess. Arch Ophthalmol. 1934;12(2):157-166.

1348

- Hatt SR, Leske DA, Castañeda YS, et al. Development of pediatric eye questionnaires for children with eye disease. *Am J Ophthalmol.* 2019;200:201-217.
- Hatt SR, Leske DA, Liebermann L, Holmes JM. Symptoms in children with intermittent exotropia and their impact on health-related quality of life. *Strabismus*. 2016;24(4):139-1344
- Hatt SR, Leske DA, Liebermann L, Mohney BG, Holmes JM. Variability of angle of deviation measurements in children with intermittent exotropia. *J AAPOS*. 2012;16(2):120-124.

IXT7ProtV1.0 19Apr2022 